# **CLINICAL STUDY PROTOCOL**

**PRODUCT:** BAX 855 – Pegylated full-length recombinant factor VIII

**STUDY TITLE:** Phase 3, prospective, randomized, multi-center clinical study comparing the safety and efficacy of BAX 855 following PK-guided prophylaxis targeting two different FVIII trough levels in subjects with severe Hemophilia A

**STUDY SHORT TITLE:** BAX 855 PK-guided Dosing

**PROTOCOL IDENTIFIER: 261303** 

**CLINICAL TRIAL PHASE 3** 

**AMENDMENT 2: 2015 MAY 12** 

Replaces:

**AMENDMENT 1: 2015 MAR 20** 

**ALL VERSIONS:** 

**AMENDMENT 2: 2015 MAY 12** 

**AMENDMENT 1: 2015 MAR 20** 

ORIGINAL: 2015 JAN 13

OTHER ID(s)

**NCT Number:** To be Determined

**EudraCT Number:** To be Determined

**IND NUMBER:** To be Determined

**Study Sponsor(s):** 

Baxalta US Inc.

**Baxalta Innovations GmbH** 

One Baxter Way

Industriestrasse 67

Westlake Village, CA 91362

A-1221 Vienna, AUSTRIA

# 1. STUDY PERSONNEL

# 1.1 Study Organization

The name and contact information of the responsible party and individuals involved with the study (eg, investigator(s), sponsor's medical expert and study monitor, sponsor's representative(s), laboratories, steering committees, and oversight committees [including ethics committees (ECs)], as applicable) will be maintained by the sponsor and provided to the investigator.

#### 2. SERIOUS ADVERSE EVENT REPORTING

The investigator will comply with applicable laws/requirements for reporting serious adverse events (SAEs) to the ECs.

# ALL SAEs ARE TO BE REPORTED ON THE SERIOUS ADVERSE EVENT REPORT (SAER) FORM AND TRANSMITTED TO THE SPONSOR WITHIN 24 HOURS AFTER BECOMING AWARE OF THE EVENT

See SAER form for contact information.

Further details are also available in the study team roster.

For definitions and information on the assessment of these events, refer to the following:

- AE, Section 13.2
- SAE, Section 13.2.1.1
- Assessment of AEs, Section 13.2.2

#### 3. SYNOPSIS

| INVESTIGATIONAL PRODUCT | |
|---|---|
| Name of Investigational<br>Product (IP) | BAX 855 |
| Name(s) of Active Ingredient(s) | Pegylated full-length Recombinant Factor VIII |
| CLINICAL CONDITION(S)/INDICATION(S) | |
| • Treatment and prophylaxis of bleeding in severe Hemophilia A | |
| PROTOCOL ID | 261303 |
| PROTOCOL TITLE | Phase 3, prospective, randomized, multi-center clinical study comparing the safety and efficacy of BAX 855 following PK-guided prophylaxis targeting two different FVIII trough levels in subjects with severe Hemophilia A |
| Short Title | BAX 855 PK-Guided Dosing |
| STUDY PHASE | Ph3 |
| PLANNED STUDY PERIOD | |
| Initiation | First subject in: Q3 2015 |
| Primary Completion | Q4 2017 |
| Study Completion | Q2 2018 |
| Duration | 3 years |
| STUDY OR IFCTIVES AND DUDDOSE | |

#### STUDY OBJECTIVES AND PURPOSE

#### **Study Purpose**

- 1. To compare the efficacy and safety of PK-guided treatment with BAX 855 targeting FVIII trough levels of 1-3% and approximately 10% (8-12%)
- 2. To further characterize pharmacokinetic (PK) and pharmacodynamic (PD) parameters of BAX 855

# **Primary Objective**

1. The primary objective is to compare two prophylactic dosing regimens of BAX 855 targeting two different FVIII trough levels, by comparing the proportions of subjects achieving a total annualized bleeding rate (ABR) of 0 in the second 6-month study period

#### **Secondary Objectives**

The secondary objectives are

- To compare the two prophylactic dosing regimens of BAX 855 targeting two different FVIII trough levels with respect to the following:
  - ➤ The proportion of subjects in each prophylactic dosing arm achieving a spontaneous ABR and spontaneous i joint bleeding rate (AJBR) of 0 in the second 6-month study period
  - The proportion of subjects in each prophylactic dosing arm with a total, spontaneous ABR and AJBR <2

i.e. not trauma related.

- ➤ The total, spontaneous, and trauma-related ABRs in the 12-month study period
- > The reduction in ABR between the two treatment arms and the historical ABR prior to study enrollment
- The total weight-adjusted consumption of BAX 855 for each prophylactic regimen
- > The joint status using the Hemophilia Joint Health Score (HJHS) and over time
- > The pharmacoeconomic outcomes
- To determine the hemostatic efficacy of BAX 855 in the control of bleeding episodes
- To evaluate the efficacy of BAX 855 for perioperative management, if surgery is required
- To determine the immunogenicity of BAX 855
- To determine the safety of BAX 855
- To determine the PK parameters of BAX 855 at baseline and steady state and the correlation with pre-infusion VWF antigen level
- To determine IR over time
- To assess the difference in the SF-36 physical domain and component change scores from baseline to follow-up between patients in the 10% trough arm and patients in the 1-3% trough arm
- To assess the difference in the change of days of physical activity participation from baseline to follow-up between patients in the 10% trough arm and patients in the 1-3% trough arm

# **Exploratory objectives:**

- To determine the potential correlation between thrombin generation assay (TGA) parameters, FVIII trough levels and ABR
- To assess the change in bleed and pain severity scores as measured by the Haemo-SYM questionnaire
- To assess the change in HRQoL using EQ-5D and mental domain and component score of the SF-36
- To assess the difference in the change in healthcare resource utilization from baseline to follow-up between patients in the 10% trough arm and patients in the 1-3% trough arm

# STUDY DESIGN

| | <del>-</del> |
|---|---|
| Study Type/ | Efficacy, Pharmacokinetic, Safety including Immunogenicity, and |
| Classification/ Discipline | Pharmacodynamic |
| Control Type | Dose-Response |
| <b>Study Indication Type</b> | Prevention, Treatment |
| Intervention model | Parallel design |
| Blinding/Masking | Open label |
| Study Design | This study is a Phase 3, prospective, randomized, open-label, multicenter study to compare the safety and efficacy of a PK-guided BAX 855 treatment regimen targeting two different FVIII trough levels in approximately 116 subjects with severe hemophilia A to have 96 subjects evaluable (48 per treatment arm). |

# Planned Duration of **Subject Participation**

The subject's participation will last approximately 15-16 months and is based on the assumption that completion of screening procedures will require approximately 6 weeks; PK assessments, dose calculation and randomization will take 6-8 weeks and the treatment period from the baseline visit to study completion will be 12 months.

#### **Primary Outcome Measure**

1. Total ABR

#### **Secondary Outcome Measures**

#### Efficacy

- 1. Total, spontaneous and traumatic ABR, and spontaneous AJBR
- 2. Total weight-adjusted consumption of BAX 855
- 3. Overall hemostatic efficacy rating at 24 ( $\pm$  2) hours after the initiation of treatment and at resolution of bleed
- 4. Number of BAX 855 infusions needed for the treatment of bleeding episodes
- HJHS
- 6. Intra-, post- and perioperative hemostatic efficacy in case of surgery
- 7. Intra- and postoperative blood loss in case of surgery

#### Safety

- 1. Occurrence of AEs and SAEs
- 2. Clinically significant changes in vital signs and clinical laboratory parameters (hematology, clinical chemistry, and lipids)
- 3. Inhibitory antibodies to FVIII, and binding antibodies to FVIII, BAX 855, PEG, and CHO protein

#### **Patient Reported Outcomes (PROs)**

1. Physical domain and component scores of the SF-36 Physical activity level

#### **Pharmacokinetics**

- 1. BAX 855 PK parameters based on FVIII activity at baseline and steady state:
  - a. AUC0-∞ (Area under the plasma concentration versus time curve from time 0 to infinity), IR (incremental recovery) at 30 minutes post-infusion, T1/2 (plasma half-life), MRT (mean residence time), CL (clearance), maximum plasma concentration (Cmax) and time to maximum concentration in plasma (Tmax), Vss (Volume of distribution at steady state)
  - b. Incremental recovery (IR) over time

#### **Exploratory Outcome Measures**

- 1. Thrombin generation assay (TGA) parameters (lag time, time to peak thrombin generation, peak thrombin generation, and endogenous thrombin potential [ETP])
- 2. Bleed and pain severity scores as measured by the Haemo-SYM questionnaire
- 3. HRQoL as assessed using EQ-5D and mental domain and component scores of the SF-36
- 4. Healthcare resource utilization

| INVESTIGATIONAL PRODUCT(S), DOSE AND MODE OF ADMINISTRATION | |
|---|---|
| Active Product | BAX 855 Dosage form: injection, powder, lyophilized, for solution |
| | Dose and Dosage frequency: BAX 855 dose will be PK-guided to maintain FVIII target trough levels of 1-3% or approximately 10% (8-12%) at the following dosing frequencies: FVIII trough levels of 1-3%: approximately twice weekly <sup>ii</sup> FVIII trough levels of approximately 10% (8-12%): every other day Mode of Administration: intravenous bolus |
| SUBJECT SELECTION | |
| Targeted Accrual | Approximately 116 subjects will be enrolled to have 96 subjects evaluable (48 in each prophylaxis dosing arm). |
| Number of<br>Groups/Arms/Cohorts | 2 |

#### Inclusion Criteria for Subjects Transitioning from Another BAX 855 study:

- 1. Subject has completed the end of study visit of a BAX 855 study or is transitioning from the ongoing Continuation Study 261302
- 2. Subject is either receiving on-demand or prophylactic treatment with BAX 855 and had an ABR of ≥ 2 documented and treated during the past 12 months
- 3. Subject is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm³, as confirmed by central laboratory
- 4. Subject is willing and able to comply with the requirements of the protocol

# **Inclusion Criteria for Newly Recruited Subjects:**

- 1. Subject is 12 to 65 years old at the time of screening
- 2. Subject has severe hemophilia A (FVIII clotting activity < 1%) as confirmed by central laboratory or by historically documented FVIII clotting activity performed by a certified clinical laboratory and/or a FVIII gene mutation consistent with severe hemophilia A
- 3. Subject has been previously treated with plasma-derived FVIII concentrates or recombinant FVIII for ≥ 150 documented exposure days (EDs)
- 4. Subject is either receiving on-demand treatment or prophylactic treatment and had an annual bleeding rate of ≥ 2 documented and treated during the past 12 months.
- 5. Subject has a Karnofsky performance score of ≥ 60 at screening
- 6. Subject is HIV-; or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm³, as confirmed by central laboratory at screening
- 7. Subject is hepatitis C virus negative (HCV-) by antibody (if positive, additional PCR testing will be performed), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis
- 8. If female of childbearing potential, subject presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study
- 9. Subject is willing and able to comply with the requirements of the protocol.

\_

<sup>\*</sup>Twice weekly: infusion on day 3 or 4, at two different doses to cover the different treatment intervals, or every 3.5 days. According to individual PK, frequency may be adjusted based on FVIII trough levels.

#### **Exclusion Criteria**

#### **Exclusion Criteria for Subjects Transitioning from Another BAX 855 study:**

- Subject has developed a confirmed inhibitory antibody to FVIII with a titer of ≥ 0.6 BU using the Nijmegen modification of the Bethesda assay as determined at the central laboratory during the course of the previous BAX 855 study
- 2. Subject has been diagnosed with an acquired hemostatic defect other than hemophilia A
- 3. The subject's weight is < 35 kg or > 100 kg
- 4. Subject's platelet count is < 100,000/mL
- 5. Subject has an abnormal renal function (serum creatinine > 1.5 times the upper limit of normal)
- 6. Subject has active hepatic disease with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels  $\geq 5$  times the upper limit of normal
- 7. Subject is scheduled to receive an immunomodulating drug (eg, corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or α-interferon) other than anti-retroviral chemotherapy during the study
- 8. Subject has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject's safety or compliance
- 9. Subject is planning to take part in any other clinical study during the course of the study, with the exception of BAX 855 Surgery Study as described in this protocol
- 10. Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study

# **Exclusion Criteria for Newly Recruited Subjects**

- 1. Subject has detectable FVIII inhibitory antibodies ( $\geq 0.6~BU$  using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening
- Subject has a history of confirmed FVIII inhibitors with a titer ≥ 0.6 Bethesda Units (BU) (as
  determined by the Nijmegen modification of the Bethesda assay or the assay employed with the
  respective cut-off in the local laboratory) at any time prior to screening
- 3. Subject has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease)
- 4. The subject's weight is < 35 kg or > 100 kg.
- 5. Subject's platelet count is < 100,000/mL.
- 6. Subject has known hypersensitivity towards mouse or hamster proteins, PEG or Tween 80
- 7. Subject has severe chronic hepatic dysfunction [eg, ≥ 5 times upper limit of normal alanine aminotransferase (ALT) and/ or aspartate aminotransferase (AST), as confirmed by central laboratory at screening, or a documented INR > 1.5]
- 8. Subject has severe renal impairment (serum creatinine > 1.5 times the upper limit of normal)
- 9. Subject has current or recent (< 30 days) use of other pegylated drugs prior to study participation or is scheduled to use such drugs during study participation
- 10. Subject is scheduled to receive during the course of the study, a systemic immunomodulating drug (eg, corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or  $\alpha$ -interferon) other than anti-retroviral chemotherapy.

- 11. Subject has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
- 12. Subject has a medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance
- 13. Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

#### STATISTICAL ANALYSIS

#### **Sample Size Calculation**

For the sample size assessment the following assumptions were used: Approximately 40% of patients in BAX 855 regimen targeting 1-3% trough level are expected to be bleed free as shown in the ADVATE Prophylaxis study and the BAX 855 pivotal study 261201. For the BAX 855 regimen targeting approximately 10% (8-12%) trough level, there are no reliable data available. However, an increase of 30% in bleed free patients is considered clinically relevant.

If the above assumptions hold true 48 subjects per study group are needed to reject the null hypothesis of no difference between the study groups with 80% power. Significance level of the test is targeted at 5% two-sided level. Assuming a drop-out rate of close to 10%, and 10-15% of subjects being non-compliant, approximately 116 subjects are planned to be randomized between the two BAX 855 regimens with an allocation ratio of 1:1.

#### **Planned Statistical Analysis**

The proportion of subjects with ABR = 0 in the two prophylaxis treatment regimens will be compared using a chi-square test with continuity correction (at a two-sided 5% level of significance). For all outcome measures, bleeding rates will be analyzed using a negative binomial model and descriptive statistics will be presented for the two dosing regimens for other outcomes. Point estimates (mean or median) and 95% CIs will be computed if feasible.

# 4. TABLE OF CONTENTS

| 1. STUDY PERSONNEL | 2 |
|-------------------------------------------------------------------|----|
| 1.1 Study Organization | 2 |
| 2. SERIOUS ADVERSE EVENT REPORTING | 3 |
| 3. SYNOPSIS | 4 |
| 4. TABLE OF CONTENTS | 10 |
| 5. LIST OF ABBREVIATIONS | 15 |
| 6. BACKGROUND INFORMATION | 18 |
| 6.1 Description of Investigational Product | 18 |
| 6.2 Clinical Condition/Indication | |
| 6.3 Population To Be Studied | 20 |
| 6.4 Findings from Nonclinical and Clinical Studies | |
| 6.4.1 Findings from Nonclinical Studies | |
| 6.4.2 Findings from Clinical Studies | |
| 6.5 Evaluation of Anticipated Risks and Benefits of the Investiga | |
| Human Subjects | |
| 6.6 Authorized Representative (Signatory) / Responsible Party | |
| 6.7 Compliance Statement | 20 |
| 7. STUDY PURPOSE AND OBJECTIVES | 27 |
| 7.1 Study Purpose | 27 |
| 7.2 Primary Objective | |
| 7.3 Secondary Objectives | |
| 7.3.1 Efficacy | 27 |
| 7.3.2 Safety | |
| 7.3.3 Pharmacokinetics | |
| 7.3.4 Patient Reported Outcomes | |
| 7.4 Exploratory Objectives | 28 |
| 8. STUDY DESIGN | 29 |
| 8.1 Brief Summary | 29 |
| 8.2 Overall Study Design | |
| 8.3 Duration of Study Period(s) and Subject Participation | |
| 8.4 Outcome Measures | |
| 8.4.1 Primary Outcome Measure | |

| 8.4.2 Secondary Outcome Measures | 30 |
|---|---|
| 8.4.2.1 Efficacy | 30 |
| 8.4.2.2 Safety | 31 |
| 8.4.2.3 Patient Reported Outcomes | |
| 8.4.2.4 Pharmacokinetics | |
| 8.4.3 Exploratory Outcome Measures | |
| 8.5 Randomization and Blinding | |
| 8.6 Study Stopping Rules | |
| 8.7 Investigational Product(s) | |
| 8.7.1 Packaging, Labeling, and Storage | |
| 8.7.2 Administration | |
| 8.7.3 Description of Treatment | 33 |
| 8.7.3.1 BAX 855 Dosing for PK Assessment | |
| 8.7.3.2 BAX 855 Prophylaxis Dosing | |
| 8.7.3.3 BAX 855 Dose and/or Frequency Adjustments | |
| 8.7.3.4 Treatment of Bleeding Episodes | |
| 8.7.3.5 Treatment for Surgery or Dental Procedures | |
| 8.7.3.6 Immune Tolerance Induction for Inhibitor Development | |
| 8.7.4 Investigational Product Accountability | |
| 8.8 Source Data | |
| 9. SUBJECT SELECTION, WITHDRAWAL, AND DISCONTINUATION 9.1 Inclusion Criteria | |
| 9.1.1 Subjects Transitioning from Another BAX 855 Study | |
| 9.1.2 Inclusion Criteria for Newly Recruited Subjects | |
| 9.2 Exclusion Criteria | |
| | 41 |
| 9.2.1 Exclusion Criteria for Subjects Transitioning from Another DAA 555 | 41 |
| 9.2.1 Exclusion Criteria for Subjects Transitioning from Another BAX 855 Study | |
| Study | 41 |
| | 41<br>41 |
| Study9.2.2 Exclusion Criteria for Newly Recruited Subjects | 41<br>41 |
| Study9.2.2 Exclusion Criteria for Newly Recruited Subjects | 41<br>41<br>43 |
| Study | 41<br>41<br>43 |
| Study | 41<br>41<br>43<br>44 |
| Study | 41<br>43<br>43<br>44<br>44 |
| Study | 41<br>43<br>44<br>44<br>44<br>45 |
| Study | 41<br>43<br>44<br>44<br>44<br>45 |
| Study | 41 43 44 44 44 45 45 |
| Study | 41 43 44 44 44 45 45 45 |
| Study | 41 43 44 44 45 45 45 45 |
| Study | 41 43 44 44 45 45 45 45 45 |

| 11. ASSESSMENT OF EFFICACY | 50 |
|-------------------------------------------------------------------|----------|
| 11.1 Bleeding Assessment | 50 |
| 11.1.1 Hemostatic Efficacy Rating for Treatment of Bleeding Episo | |
| 11.1.2 Number of BAX 855 Infusions Needed for the Treatment of | |
| Episodes | |
| 11.1.3 Hemophilia Joint Health Score (HJHS) | 52 |
| 11.1.4 Weight-Adjusted Consumption of BAX 855 | 52 |
| 11.1.5 Peri-operative efficacy assessments | 52 |
| 12. DETERMINATION OF FVIII AND VWF ANTIGEN, FVIII ACTIV | VITY AND |
| TGA | 53 |
| 12.1 PHARMACOKINETICS | 53 |
| 12.2 Incremental Recovery (IR) | |
| 12.3 Trough Levels | |
| 13. ASSESSMENT OF SAFETY INCLUDING IMMUNOGENICITY | 56 |
| 13.1 Immunogenicity | 56 |
| 13.2 Adverse Events | 57 |
| 13.2.1 Definitions | 57 |
| 13.2.1.1 Serious Adverse Event | 57 |
| 13.2.1.2 Non-Serious Adverse Event | 58 |
| 13.2.1.3 Unexpected Adverse Events | |
| 13.2.1.4 Preexisting Diseases | |
| 13.2.2 Assessment of Adverse Events | |
| 13.2.2.1 Severity | |
| 13.2.2.2 Causality | |
| 13.3 Urgent Safety Measures | |
| 13.4 Untoward Medical Occurrences | |
| 13.5 Medical Device Safety reporting | |
| 13.6 Non-Medical Complaints | |
| 13.7 Medical, Medication, and Non-Drug Therapy History | |
| 13.8 Physical Examinations | |
| 13.9 Clinical Laboratory Parameters | |
| 13.9.1 Screening Laboratory Parameters | |
| 13.9.1.1 Blood Type | |
| 13.9.1.2 Genetics and HLA-Genotype | |
| 13.9.1.3 Pregnancy Test | |
| 13.9.2 CD4 Count | |
| 13.9.3 Viral Serology | |
| 13.9.4 Hematology, Clinical Chemistry and Lipid Panel | |
| 13.9.5 FVIII Activity, FVIII Antigen, VWF Antigen | |
| 13.9.6 Thrombin Generation Assay | |
| L.J.Y. / ASSESSMENT OF L'ADOCATORY VAINES | 66 |

| 15.9./.1 Assessment of Adnormal Ladoratory values | |
|-----------------------------------------------------------|----|
| 13.9.8 Biobanking | |
| 13.10 Vital Signs | 67 |
| 14. STATISTICS | 68 |
| 14.1 Sample Size and Power Calculations | 68 |
| 14.1.1 Sample Size Calculation | 68 |
| 14.2 Datasets and Analysis Cohorts | 68 |
| 14.2.1 Full Analysis Set | |
| 14.2.2 Per Protocol Analysis Set | |
| 14.2.3 Safety Analysis Set | |
| 14.3 Handling of Missing, Unused, and Spurious Data | |
| 14.3.1 Handling of incomplete observation periods for ABR | |
| 14.3.2 Handling of other variables | |
| 14.4 Methods of Analysis | |
| 14.4.1 Primary Outcome Measure | |
| 14.4.2 Secondary Outcome Measures | |
| 14.4.3 Exploratory Outcome Measures | 72 |
| 15. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 73 |
| 16. QUALITY CONTROL AND QUALITY ASSURANCE | 74 |
| 16.1 Investigator's Responsibility | |
| 16.1.1 Final Clinical Study Report | |
| 16.2 Training | |
| 16.3 Monitoring | |
| 16.4 Auditing | 74 |
| 16.5 Non-Compliance with the Protocol | |
| 16.6 Laboratory and Reader Standardization | |
| 17. ETHICS | 76 |
| 17.1 Subject Privacy | 76 |
| 17.2 Ethics Committee and Regulatory Authorities | |
| 17.3 Informed Consent | |
| 17.4 Data Monitoring Committee | |
| 18. DATA HANDLING AND RECORD KEEPING | 78 |
| 18.1 Confidentiality Policy | 78 |
| 18.2 Study Documentation and Case Report Forms | |
| 18.3 Document and Data Retention. | |
| 19. FINANCING AND INSURANCE | 79 |
| 1 / P | |

| 20. PUBLICATION POLICY | 79 |
|------------------------------------------------------------------------|-----|
| 21. SUPPLEMENTS | 80 |
| 21.1 Study Flow Charts | 80 |
| 21.2 Detailed Flow Diagram of Study Procedures | |
| 21.3 Schedule of Study Procedures and Assessments | |
| 21.4 Clinical Laboratory Assessments | |
| 22. PERIOPERATIVE MANAGEMENT | 96 |
| 22.1 Dosing Schedule and requirements for major surgery | 96 |
| 22.1.1 General | |
| 22.1.2 Preoperative and Loading Dose | |
| 22.1.3 Postoperative Dosing | |
| 22.2 Efficacy assessment | |
| 22.2.1 Intra-, Post-, and Perioperative Hemostatic Efficacy | |
| 22.2.2 Intra- and Postoperative Blood Loss | 101 |
| 23. DEFINITIONS | 102 |
| 23.1 Joint Bleeds | 102 |
| 23.2 Muscle Bleeds | 102 |
| 24. REFERENCES. | 103 |
| 25. SUMMARY OF CHANGES | 107 |
| Tables | |
| Table 1 BAX 855 Treatment Guidelines for Bleeding Episodes | 37 |
| Table 2 Efficacy Rating Scale for Treatment of Bleeding Episodes | |
| Table 3 PK Time Points | 53 |
| Table 4 IR Time Points | |
| Table 5 Intraoperative Efficacy Assessment Scale | |
| Table 6 Postoperative Efficacy Assessment Scale (Postoperative Day 1) | |
| Table 7 Perioperative Efficacy Assessment Scale (at discharge or 14 da | |
| whichever is first) | 101 |
| Figures | |
| Figure 1 Study Design for Baxalta Clinical Study 261303 | 80 |
| Figure 2 Study Flow Chart | 81 |
| Figure 3 Dosing Recommendations for Major Surgeries | |

# **5. LIST OF ABBREVIATIONS**

| Abbreviation | Definition |
|---|---|
| ABR | annualized bleeding rate |
| AE | adverse event |
| AJBR | annualized joint bleeding rate |
| ALT | alanine aminotransferase (SGPT) |
| AST | aspartate aminotransferase (SGOT) |
| AUC | area under the curve |
| AUC(0-∞) | area under the plasma concentration curve from 0 to infinity |
| BAX 855 | product code name for Baxalta's pegylated recombinant FVIII (rFVIII) |
| BU | Bethesda unit |
| (US) CFR | (US) Code of Federal Regulations |
| СНО | Chinese hamster ovary |
| CI | confidence interval |
| CL | total body clearance |
| Cmax | maximum plasma concentration |
| (e)CRF | (electronic) case report form |
| DI | dose intensification |
| DMC | data monitoring committee |
| EC | ethics committee |
| ED | exposure day |
| ELISA | enzyme-linked immunoabsorbent assay |
| EMA | European Medicines Agency |
| EQ-5D | EuroQol-5 dimension |
| ETP | endogenous thrombin potential |
| FAS | full analysis set |
| FVIII | factor VIII |
| GCP | Good Clinical Practice |
| GEE | general estimating equation |
| GLM | general linear model |
| Н | hour(s) |
| HAV | hepatitis A virus |
| HBcAb | hepatitis B core antibody |
| HBsAb | hepatitis B surface antibody |

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HCV Ab | hepatitis C virus antibody |
| HDL | high density lipoprotein |
| HIV | human immunodeficiency virus |
| НЈНЅ | hemophilia joint health score |
| HRQoL | health-related quality of life |
| IB | investigator's brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IgA | immunoglobulin A |
| IgE | immunoglobulin E |
| IgG | immunoglobulin G |
| IgM | immunoglobulin M |
| INR | international normalized ratio |
| IP | investigational product |
| IR | incremental recovery over time |
| ITI | immune tolerance induction |
| IU | international unit (s) |
| i.v. | intravenous(ly) |
| LDL | low density lipoprotein |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRT | mean residence time |
| NMC | non-medical complaint |
| PCR | polymerase chain reaction |
| PD | pharmacodynamic |
| pdFVIII | plasma-derived factor VIII |
| PEG | polyethylene glycol |
| PK | pharmacokinetic(s) |
| PKFAS | pharmacokinetic full analysis set |
| PP | per protocol |
| PPAS | per protocol analysis set |

| Abbreviation | Definition |
|------------------|-----------------------------------------|
| PRO | patient reported outcomes |
| PTP | previously treated patient |
| rFVIII | recombinant factor VIII |
| SAE | serious adverse event |
| SAER | serious adverse event report |
| SD | standard deviation |
| SF-36 | Short form-36 questionnaire |
| SIC | subject identification code |
| SWFI | sterile water for injection |
| T <sub>1/2</sub> | half-life |
| TGA | thrombin generation assay |
| Tmax | time to maximum concentration in plasma |
| US | United States |
| VAS | visual analog scale |
| VLDL | very low density lipoprotein |
| Vss | volume of distribution at steady state |
| VWF | von Willebrand factor |

#### 6. BACKGROUND INFORMATION

# 6.1 Description of Investigational Product

The investigational product (IP), BAX 855, is a polyethylene glycol (peg)-ylated full-length recombinant FVIII (rFVIII), intended for use as a FVIII replacement therapy with an extended half-life in the prophylaxis and treatment of bleeding episodes in patients with severe hemophilia A.

Since the half-life of current FVIII products is in the range of 10-14 hours <sup>1;2</sup>, current prophylaxis regimens call for infusion of FVIII every other day or every 2-3 days when based on each patient's individual PK profile.<sup>3</sup> pegylation of FVIII is designed to prolong the half-life of FVIII, with the intent of reducing the frequency of administration while maintaining similar therapeutic benefit as existing FVIII products; improving patient convenience and compliance with therapy; and thereby improving overall health outcomes. Prolongation of half-life of FVIII may also increase efficacy by increasing the FVIII trough levels while maintaining the frequency of administration of existing FVIII concentrates every other day.

BAX 855 consists of rFVIII protein molecules with covalently bound PEG chains linked to the protein using a stable linker. The product is reconstituted with sterile water for injection (SWFI) and is administered intravenously (i.v.) as a solution by bolus infusion. It uses the same stabilizing agents (mannitol, trehalose, histidine and glutathione) as the rFVIII product (octocog alfa, ADVATE) from which it is derived. Comprehensive preclinical studies as well as two successfully completed studies (Baxter clinical study 261101 and 261201) have shown that the pegylation extends both the *in vivo* half-life and the measurable circulating activity of the product (as determined by chromogenic and 1-stage clotting assays). Physiochemical characterization studies demonstrate that the functional activity of BAX 855 is comparable to that of ADVATE. Additional details can be found in the BAX 855 Investigator's Brochure (IB).

No comparator drug product will be used in this study for prophylaxis or treatment of bleeding. Treatment regimens are based on individual PK parameters and FVIII trough levels with a target trough level of 1-3% given twice weekly, or approximately 10% (8-12%) FVIII given every other day.

#### 6.2 Clinical Condition/Indication

Hemophilia A is an X-chromosome-linked recessive, congenital bleeding disorder caused by deficient or defective coagulation due to deficiency of FVIII. The absence of FVIII leads to 'spontaneous' bleeding episodes (occurring primarily in joints, muscles, and less commonly, in soft tissues) and to excessive bleeding following trauma or injury. Hemophilia A is currently treated with FVIII replacement using either plasma-derived (pdFVIII) or rFVIII concentrates. 4;5

The intended indication for BAX 855 is treatment and prophylaxis of bleeding in subjects with hemophilia A. The clinical program of BAX 855 is in compliance with the EMA/CHMP/BPWP/144533/2009 guidelines for FVIII in hemophilia A.<sup>6</sup>

The major objective of a prophylactic treatment in severe hemophilia A patients is to prevent bleeding episodes, in particular frequent joint bleeding. Bleeding episodes in a joint cause detrimental changes in synovial tissue and cartilage, which trigger synovial cell inflammation and proliferation, cartilage damage and bone erosion. Intra-articular bleeding is the most important risk factor and seems to play a key role not only for the inflammation but also for the direct destructive process in the joint. A number of prospective and retrospective clinical studies have demonstrated that prophylactic treatment reduced the number of break-through bleeds compared to on-demand treatment. 9;10;11;12;13;14;15;16;17;18

Current management of severe hemophilia A includes on-demand treatment for bleeding episodes and prophylaxis to prevent bleeds. <sup>19;20</sup> A prospective clinical study using individually pharmacokinetic (PK) adjusted prophylaxis dosing targeting a FVIII trough level of 1% can reduce the annualized bleed rate (ABR) from 44 during on demand treatment to 1 during standard prophylaxis. The optimal prophylaxis regimen is still under scientific discussion but the frequency of break through bleedings during prophylactic treatment is assumed to depend on the time spent with a low FVIII level. Thus, dose recommendations used in prophylaxis are designed to keep the FVIII trough level above 1% of the normal level. <sup>21</sup>

However, the 1% level is not applicable to prevent bleeding episodes in all patients. Especially patients with damaged joints often bleed in spite of maintenance of a 1% trough level, although this association is difficult to access in clinical practice. A pioneering bench mark study by Den Uijl et al. has suggested that the annual number of bleeds is approaching zero when baseline levels of FVIII > 10% are maintained. Association is difficult to access in clinical practice.

Although there are no established criteria for determining how many joint bleeds can be tolerated before irreversible damage occurs, some studies reported that more than 2-5 joint bleeds in total lead to impaired joint scores <sup>24;25;26</sup> whereas annual bleed rates between 0.1 and 2.7 did not lead to joint damage. <sup>27;28;29</sup>

In an advanced stage these events accumulate and result in permanent loss of joint mobility leading to crippling arthropathy, the hallmark of advanced severe hemophilia A. For the assessment of joint impairment, joint scores have been developed. One of the best established scores is the Hemophilia Joint Health Score (HJHS). The HJHS is a validated 11-item scoring tool based on radiologic and clinical evaluation, sensitive to detect early signs and minor changes. <sup>30</sup>

# 6.3 Population To Be Studied

Adolescent and adult subjects (aged 12 - 65 years) with severe hemophilia A (FVIII < 1%), of all races and ethnic groups, without history of or currently confirmed FVIII inhibitors ( $\geq 0.6$  BU) will be studied. All subjects will have been previously treated with pdFVIII or rFVIII concentrates with  $\geq 150$  documented exposure days (EDs) (previously treated patients; PTP). Subjects receiving prophylaxis and on-demand treatment will be included in this study and they must have had at least 2 documented and treated bleeds within the 12 months prior to enrolment.

Justification for enrollment of adolescent subjects is based on the nonclinical safety requirements outlined in the ICH M3 Guideline, Section 12 as well as the ICH E11 Guideline on clinical investigation of medicinal products in the pediatric population. Hemophilia is a serious and potentially life-threatening disease. Adolescent subjects, in particular if they are physically active, are expected to benefit from a new treatment approach with target FVIII trough levels of approximately 10% using a new recombinant full-length rFVIII molecule with an extended half-life. Moreover, results from nonclinical repeated toxicology studies, the core safety pharmacology package and the completed clinical phase 1 and phase 2/3 pivotal study have not raised any safety or tolerability concerns. Furthermore, the parent protein molecule ADVATE has been used extensively in the entire pediatric population with no unforeseen adverse events (AEs) (see ADVATE Company Core data Sheet).

# 6.4 Findings from Nonclinical and Clinical Studies

# **6.4.1 Findings from Nonclinical Studies**

BAX 855 is manufactured by covalently binding a branched PEG reagent with a molecular weight of 20 kDA to Baxalta's rFVIII (octocog alfa, ADVATE). Baxalta's octocog alfa is expressed in Chinese hamster ovary (CHO) cells by a plasma/albumin free cell culture method and is the active substance in Baxalta's licensed product ADVATE. Thus, the viral safety of BAX 855 is ensured by the octocog alfa (ADVATE) bulk drug substance manufacturing process as any potential risk of contamination with viruses or adventitious agents during the subsequent manufacturing steps of BAX 855 has been minimized. No substances of animal or human origin are added throughout the entire manufacturing process of BAX 855.

Preclinical studies have demonstrated BAX 855 to have comparable activity and other biochemical properties to ADVATE. The expected prolonged FVIII exposure by BAX 855 was demonstrated in PK studies with a mean residence time (MRT) longer than ADVATE in FVIII knock-out-mice (1.6 fold), rats (1.2 fold) and cynomolgus monkeys (1.5 fold). Prolonged efficacy was shown for BAX 855 in comparison to equivalent doses of ADVATE in two primary pharmacodynamic models in FVIII knock-out mice.

Additional data from nonclinical studies can be found in the BAX 855 IB.

# **6.4.2 Findings from Clinical Studies**

A Phase 1, first in human study (Baxter clinical study 261101) to assess the safety and PK of BAX 855 in PTPs aged 18-65 years with severe hemophilia A with ≥150 EDs to FVIII products was conducted in Europe and Japan. The study investigated safety and PK of single doses of 30 IU/kg and 60 IU/kg BAX 855 compared to the same dose of ADVATE. Subjects were followed for 28 days after BAX 855 administration for safety. Safety assessments included AEs, changes in vital signs, clinical laboratory assessments, and immunogenicity.

A total of 24 subjects were enrolled; 19 were treated and 18 were evaluable for PK analysis. Nine were treated with 30 IU/kg (Cohort 1) and 10 were treated with 60 IU/kg (Cohort 2) of BAX 855, including 2 subjects from Japan.

No subjects developed inhibitors to FVIII or binding antibodies to PEG after BAX 855 infusion. Binding antibodies to FVIII and PEG-FVIII were present in some subjects after BAX 855 infusion but all were at the lowest detectable titers (ie, 1:20 or 1:40); these results could not be analyzed for specificity and were therefore interpreted as "low-titer indeterminate". Furthermore, no increases in preexisting antibody titers were observed after BAX 855. There were no thrombosis-associated events or allergic reactions.

No deaths or other serious adverse events (SAEs) occurred, and none of the 11 non-serious AEs (all mild or moderate) were considered treatment-related. AEs reported following BAX 855 administration included vomiting, nasopharyngitis, upper respiratory tract infection, influenza-like illness, arthralgia, headache, and localized swelling. No significant treatment-related changes in laboratory values or vital signs were recorded. There were no notable differences in the type or rate of AEs experienced by subjects after ADVATE infusion versus BAX 855 infusion.

Eighteen subjects (Cohort 1, n=8; Cohort 2, n=10) were evaluable for PK analysis. Based on the one-stage clotting assay, the median elimination phase half-life ( $T_{1/2}$ ; h) was longer for BAX 855 than for ADVATE in both Cohort 1 (13.60 vs 9.90) and Cohort 2 (16.64 vs 11.11). Other PK parameters also supported an improved PK profile for BAX 855 compared to ADVATE. Refer to the ADVATE Company Core Data Sheet for more details on the clinical experience to date with ADVATE.

Based on these data, BAX 855 appears to be safe and well tolerated after a single dose administration. The mean  $T_{1/2}$  was 1.4 and 1.5-fold higher for BAX 855 compared to ADVATE in Cohorts 1 and 2, respectively, demonstrating prolonged circulation of BAX 855 compared to ADVATE. These data support the use of the BAX 855 dosing regimens planned in this study.

In phase 2/3 study 261201, BAX 855 was found to be safe and well tolerated in all 137 treated subjects, with an accumulated total of 6717 EDs to BAX 855 and 21,803,981 IU of BAX 855 infused. None of the subjects developed inhibitory antibodies to FVIII of ≥ 0.6 BU/mL or persistent binding antibodies to FVIII, PEG-FVIII or PEG. No subjects developed antibodies to CHO proteins. Binding antibodies that were detected prior to exposure to BAX 855 or that transiently developed during the study could not be correlated to an impaired treatment efficacy, altered PK parameter, or temporally associated AE. Based on these data, no increased risk for PTPs with ≥150 EDs to develop inhibitory antibodies to FVIII, no immune responses with a clinical impact, and no evidence of allergic or hypersensitivity reactions were observed in this study.

Seven adverse reactions including headache, diarrhea, nausea, and flushing occurred in 6 subjects. All adverse reactions were consistent with the pharmacology of ADVATE. There were no allergic reactions or deaths related to BAX 855 during the study. Although some changes were observed in laboratory assessments for liver enzymes (alanine aminotransferase (ALT) and aspartate aminotransferase (AST)) these were attributed to preexisting disease, in particular to hepatitis C virus (HCV) infection. There were no related SAEs and no safety signals were observed during the study.

PK parameters of BAX 855 and ADVATE at the same dose level in dose-escalation study 261101 and in the pivotal study 261201 suggest that pegylation offers prolonged circulating FVIII levels in subjects with severe hemophilia A. Duration of circulation at the 30 IU/kg, 45 IU/kg, and the 60 IU/kg dose level was longer for BAX 855 than for ADVATE. In addition, the PK profile demonstrated that AUC0-∞ increases proportionally with increasing dose levels.

In study 261201, at a prophylactic dose level of  $45 \pm 5$  IU/kg, the estimated mean fold increase with BAX 855 compared to ADVATE was approximately 1.4-fold for  $T_{1/2}$ , approximately 1.5-fold for MRT, and approximately 1.9-fold for AUC0- $\infty$  in the one-stage clotting assay. Fold increases in PK parameters were consistent in adolescent and adult subjects. Using the chromogenic assay, fold increases were similar for the pegylated extended half-life product compared to the licensed rFVIII product. BAX 855 PK outcomes remained consistent between the initial and repeat PK infusions after  $\geq$ 50 EDs indicating that repeated exposure did not affect the PK profile of BAX 855.

In terms of efficacy, study 261201 met its primary endpoint by demonstrating a reduction of the mean ABR for prophylaxis of more than 50% compared to on-demand treatment using a negative binomial model analysis as determined in the full analysis set (FAS) of all subjects who received BAX 855 for prophylaxis or on-demand. The ratio for the mean ABR for prophylaxis to the mean ABR for on-demand treatment was 0.10 (95% CI 0.06; 0.19); the estimated mean ABRs were 4.3 (95% CI: 3.4; 5.5) for prophylaxis and 43.4 (95% CI: 25.2; 74.8) for on-demand treatment with BAX 855. An analysis by age group was not feasible for the adolescents due to the small number of subjects in the on-demand treatment group (n=2), however, subjects aged 18 to 65 years demonstrated similar mean ABRs to the overall group and a statistically significant reduction in ABR for prophylaxis compared to on-demand treatment.

A mean (SD) of 1.86 (0.31) and a median (Q1; Q3) of 1.96 (1.89; 1.99) prophylactic infusions per week were administered at a dose of mean (SD) of 44.36 (3.88) IU/kg and a median (95% CI) of 44.83 (44.19; 45.43) IU/kg dose per infusion, suggesting that the subjects in the study received BAX 855 for prophylaxis twice weekly at  $45 \pm 5$  IU/kg as intended according to the protocol.

A total of 39.6% (40/101) of subjects in the per protocol analysis set (PPAS) who were treated with their originally assigned prophylactic dose for the entire duration of study participation and who fulfilled pre-specified compliance requirements, had zero bleeding episodes, none (0/17) of the subjects in the on-demand arm was bleed-free.

In the prophylaxis arm, 57.4% (58/101) of subjects had no spontaneous bleeding episodes and 57.4% (58/101) had no joint bleeding episodes.

The intervals between bleeding episodes were longer for subjects on prophylaxis than those treated on-demand (PPAS): 15.8% (16/101) of subjects on prophylaxis had  $\leq 1$  month between bleeding episodes compared with 100% (17/17) of subjects treated on demand.

Descriptive statistics reflecting the PPAS demonstrated a lower median (Q1; Q3) ABR (1.9 [0.0; 5.8]) in the prophylaxis arm (n = 101) compared to the on-demand arm (41.5 [31.7; 51.1]; n = 17) for all bleeding episodes.

These results demonstrate that BAX 855 used at the intended infusion interval and dose is efficacious in the reduction of the ABR in PTPs with severe hemophilia A compared to on-demand treatment.

BAX 855 was also efficacious in the treatment of bleeding episodes. The pre-defined success rate at 24 h as assessed by the proportion of subject with bleeds (n = 70) rated excellent or good on a 4-point scale was 0.97 (95% CI 0.94; 0.98) which was significantly higher (p <0.0001) than the null hypothesis of a success rate of 70% which was considered to be the lowest clinically acceptable success rate.

Hemostatic efficacy at 24 hours after infusion was rated excellent or good in >90% of bleeding episodes across bleeding sites (joint and non-joint) and etiologies (spontaneous/unknown and injury-related). Across bleeding sites and etiologies, >90% of all bleeding episodes in the PPAS were treated with only 1 or 2 infusions.

Physical activity level participation was collected as an exploratory outcome measure in the pivotal trial and analyzed post hoc for patients who were previously on-demand and then switched to prophylaxis with BAX 855 in the study. These patients (n=18) demonstrated an increase in their mean days of activity of 3.06 days per week (SD:5.90) from baseline to follow-up. They also demonstrated clinically meaningful improvements in their physical health-related quality of life in the Role Physical, Bodily Pain, and Physical Component Scores.

The results of these studies demonstrate that BAX 855 is safe and efficacious in treating bleeding episodes and in prophylaxis administered twice weekly in adults and adolescents with severe hemophilia A. In addition, the data consistently demonstrate prolonged circulation of BAX 855 in comparison with the parent molecule ADVATE.

# 6.5 Evaluation of Anticipated Risks and Benefits of the Investigational Product to Human Subjects

Page 25 of 110

2015 MAY 12

BAX 855 and ADVATE have undergone comparable preclinical single and repeated dose toxicology and pharmacology testing. The results suggest that BAX 855 has a comparable safety profile to ADVATE. Since the core protein of BAX 855 is identical to ADVATE, a safety profile similar to ADVATE is expected for BAX 855 when infused in humans. The most commonly reported adverse drug reactions described for ADVATE in post-marketing clinical studies include: FVIII inhibitors, pyrexia, and headache. Allergic-type hypersensitivity reactions, including anaphylaxis, have been reported with ADVATE and have been manifested by dizziness, paresthesia, rash, flushing, face swelling, urticaria, and pruritus. iii Additional safety experience for ADVATE is provided in the ADVATE Company Core Data Sheet.

Since BAX 855 is a pegylated form of ADVATE, there is also the potential risk of inducing anti-PEG antibodies following BAX 855 administration. Binding antibodies against PEG are present in the healthy population and in patients with hemophilia A. BAX 855 may react with pre-existing anti-PEG antibodies, potentially resulting in a clinical hypersensitivity reaction or increased clearance of BAX 855 from circulation. BAX 855 and ADVATE showed a similar immunogenicity profile in preclinical in vitro and in vivo studies. Data from preclinical studies indicate that pegylated human FVIII can only induce antibodies against PEG when FVIII is recognized as a foreign protein that can provide immunogenic epitopes for CD4+ T cells. In the pivotal phase 2/3 studies it could be demonstrated that the presence of anti-PEG antibodies at screening or transiently occurring in some subjects did not have an impact on hemostatic efficacy or safety and that BAX 855 did not induce persistent antibodies to PEG or BAX 855.

Previously treated patients (PTPs) with a high degree of previous exposure to FVIII should be immunetolerant to FVIII and are considered to have a low risk of developing antibodies against FVIII. Therefore, the risk for PTPs with severe hemophilia A who do not have neutralizing antibodies against FVIII (inhibitors) are also expected to be at low risk to develop antibodies against BAX 855. In the pivotal study 261201, 101 subjects accumulated  $\geq$ 50 EDs and none of them developed inhibitory antibodies to FVIII  $\geq$  0.6 BU at any time during the study. Also, none of the subjects developed persistent binding antibodies to FVIII, PEG-FVIII or PEG. Moreover, no immune responses with a clinical impact and no evidence of hypersensitivity reactions were observed.

ADVATE Company Core Data Sheet on file at Baxalta US Inc. (Westlake Village, CA).

BAX 855 has been administered as a single dose of 30 IU/kg to 9 subjects and a single dose of 60 IU/kg to 10 subjects with severe hemophilia A in a Phase 1 study (Baxter clinical study 261101). In a Phase 2/3 study (Baxter Pivotal study 261201), the prophylactic treatment regimen of  $45 \pm 5$  IU/kg twice weekly was planned to be administered for  $\geq$  50 EDs or 6 months  $\pm$  2 weeks, whichever occurred last. On-demand therapy with BAX 855 at a dose of 10 to  $60 \pm 5$  IU/kg was to be administered for 6 months  $\pm$  2 weeks. BAX 855 was safe and well tolerated in all 137 treated subjects, with an accumulated total of 6717 EDs to BAX 855 and 21,803,981 IU of BAX 855 infused. Based on data from these two studies (see Section 6.4.2), there currently are no anticipated risks of BAX 855, beyond those associated with ADVATE, when administered in human subjects.

The comparability of BAX 855 to ADVATE, the preclinical safety profile of BAX 855, and the clinical data from the Phase 1 and 2/3 studies, suggest an acceptable risk benefit profile for BAX 855. Additional details related to risks and benefits can be found in the BAX 855 IB.

# 6.6 Authorized Representative (Signatory) / Responsible Party

PPD , MD PPD , Clinical Development Baxalta US Inc.

# **6.7 Compliance Statement**

This study will be conducted in accordance with this protocol, the International Conference on Harmonisation Guideline for Good Clinical Practice E6 (ICH GCP, April 1996), Title 21 of the US Code of Federal Regulations (US CFR), the European Clinical Trial Directive (2001/20/EC and 2005/28/EC), and applicable national and local regulatory requirements.

#### 7. STUDY PURPOSE AND OBJECTIVES

# 7.1 Study Purpose

The purpose of the study is:

- To compare the efficacy and safety of PK-guided treatment with BAX 855 targeting FVIII trough levels of 1-3% and approximately 10% (8-12%).
- To further characterize PK and PD parameters of BAX 855

# 7.2 Primary Objective

The primary objective of the study is to compare two prophylactic dosing regimens of BAX 855 targeting two different FVIII trough levels, by comparing the proportions of subjects achieving a total ABR of 0 in the second 6-month study period.

# 7.3 Secondary Objectives

# 7.3.1 Efficacy

The secondary objectives are:

- 1. To compare the two prophylactic dosing regimens of BAX 855 targeting two different FVIII trough levels with respect to the following:
  - The proportion of subjects in each prophylactic dosing arm achieving a spontaneous iv ABR and spontaneous joint bleeding rate (AJBR) of 0 in the second 6-month study period
  - The proportion of subjects in each prophylactic dosing arm with a total, spontaneous ABR and AJBR < 2
  - The total, spontaneous, and trauma-related ABRs in the 12-month study period
  - The reduction in ABR between the two treatment arms and the historical ABR prior to study enrollment
  - The total weight-adjusted consumption of BAX 855 for each prophylactic regimen
  - The joint status using the Hemophilia Joint Health Score (HJHS) and over time
  - The pharmacoeconomic outcomes
- 2. To determine the hemostatic efficacy of BAX 855 in the control of bleeding episodes

\_

iv i.e. not trauma-related

3. To evaluate the efficacy of BAX 855 for perioperative management, if surgery is required

# **7.3.2** Safety

- 1. To determine the immunogenicity of BAX 855
- 2. To determine the safety of BAX 855

#### 7.3.3 Pharmacokinetics

- 1. To determine the PK parameters of BAX 855 at baseline and steady state and the correlation with pre-infusion VWF antigen level
- 2. To determine IR over time

# 7.3.4 Patient Reported Outcomes

- 1. To assess the difference in the SF-36 physical domain and component change scores from baseline to follow-up between patients in the 10% trough arm and patients in the 1-3% trough arm
- 2. To assess the difference in the change of days of physical activity participation from baseline to follow-up between patients in the 10% trough arm and patients in the 1-3% trough arm

# 7.4 Exploratory Objectives

- 1. To determine the potential correlation between thrombin generation assay (TGA) parameters, FVIII trough levels and ABR
- 2. To assess the change in bleed and pain severity scores as measured by the Haemo-SYM questionnaire
- 3. To assess the change in HRQoL using EQ-5D and mental domain and component scores of the SF-36
- 4. To assess the difference in the change in healthcare resource utilization from baseline to follow-up between patients in the 10% trough arm and patients in the 1-3% trough arm

#### 8. STUDY DESIGN

# 8.1 Brief Summary

This study is a Phase 3, prospective, randomized, open-label, multicenter study to compare the safety and efficacy of a PK-guided BAX 855 treatment regimen targeting two different FVIII trough levels of 1-3% and approximately 10% (8-12%) in adolescent and adult PTPs with severe hemophilia A (<1% FVIII). Enrolled subjects will undergo an initial PK assessment following a single administration of BAX 855 to determine the subject's individual PK parameters to tailor the dose for the targeted FVIII trough levels. Subjects will be randomized to one of 2 study arms of 58 subjects each, to target trough FVIII levels of 1-3% or approximately 10% (8-12%), for a treatment period of 12 months. Repeat PK at steady state will be performed after 9 months of treatment.

# 8.2 Overall Study Design

This study is a Phase 3, prospective, randomized, open-label, multicenter study to compare the safety and efficacy of PK and FVIII trough level-guided BAX 855 treatment targeting FVIII trough levels of 1-3% or approximately 10% (8-12%) in a total of 96 evaluable (48 in each of two study arms) adolescent and adult PTPs with severe hemophilia A (<1% FVIII). Approximately 116 subjects will be enrolled for a total of 96 evaluable subjects (assuming a dropout rate of close to 10% and 10-15% of subjects being non-compliant). Subjects from the BAX 855 continuation (261302) the BAX 855 surgery (261204) study, the BAX 855 pediatric (261202) study, and newly recruited subjects including BAX 855-naïve subjects will participate.

Subjects will be screened per protocol inclusion/exclusion criteria and, following confirmation of eligibility, will undergo an initial PK assessment following a single administration of BAX 855 ( $60 \pm 5$  IU/kg) to determine PK parameters. Following the PK assessment subjects will be randomized to one of 2 dosing regimens: The standard treatment arm with twice weekly dosing will target FVIII trough levels of 1-3% and the second, intensified treatment arm with dosing every other day will target trough level of approximately 10% (8-12%) FVIII. The dose will be based on each subject's individual PK. More frequent dosing should be considered if single doses of 80 IU/kg are required or regular FVIII peak levels of 200 % would be reached.

Subjects will complete study visits as follows to undergo efficacy, safety, and PRO assessments: Baseline Visit, Visit 1 at 4 weeks  $\pm$  5 days; Visit 2 at 8 weeks  $\pm$  1 week; Visit 3 at 3 months  $\pm$  2 weeks; Visit 4 at 4.5 months  $\pm$  2 weeks; Visit 5 at 6 months

<sup>&</sup>lt;sup>v</sup> In case subject is at least 12 years of age at the time of informed consent of this study.

 $\pm$  2 weeks; Visit 6 at 7.5 months  $\pm$  2 weeks; Visit 7 at 9 months  $\pm$  2 weeks; Visit 8 at 10.5 months  $\pm$  2 weeks; and the Study Completion/Termination Visit for follow-up at 12 months  $\pm$  2 weeks. The following items are discussed with the subject: concomitant medications, non-drug therapies, adverse events, bleeding episodes and their treatment, including details of target joint bleedings, and to review the subject diary. For subjects without bleeding episodes, Visits 6 and 8 are phone visits. If, however, a subject has a bleeding episode, instead of a phone visit the subject must attend a site visit to assess FVIII trough levels and IR and re-evaluate the PK-guided regimen, the subject's physical activity and compliance. In these cases the subject will undergo all planned assessments for a study visit, including assessment of vital signs, physical examination, and all laboratory assessments.

The overall study design is illustrated in Figure 1.

# 8.3 Duration of Study Period(s) and Subject Participation

The overall duration of the study is approximately 3 years from study initiation (ie, first subject enrolled) to study completion. The recruitment period is expected to be approximately 15 months.

The subject participation period is approximately 15 to 16 months from enrollment to subject completion (ie, last study visit), unless prematurely discontinued.

#### **8.4 Outcome Measures**

#### **8.4.1 Primary Outcome Measure**

The primary outcome measure is the total ABR.

# **8.4.2 Secondary Outcome Measures**

# **8.4.2.1** Efficacy

- 1. Total, spontaneous and traumatic ABR, and spontaneous AJBR
- 2. Total weight-adjusted consumption of BAX 855
- 3. Overall hemostatic efficacy rating at  $24 \pm 2$  hours after the initiation of treatment and at resolution of bleed
- 4. Number of BAX 855 infusions needed for the treatment of bleeding episodes
- 5. HJHS
- 6. Intra-, post- and perioperative hemostatic efficacy in case of surgery
- 7. Intra- and postoperative blood loss in case of surgery

# 8.4.2.2 Safety

- 1. Occurrence of AEs and SAEs
- 2. Clinically significant changes in vital signs and clinical laboratory parameters (hematology, clinical chemistry, and lipids)
- 3. Inhibitory antibodies to FVIII, and binding antibodies to FVIII, BAX 855, PEG, and CHO protein

# **8.4.2.3 Patient Reported Outcomes**

1. Physical domain and component scores of the SF-36Physical activity level

#### 8.4.2.4 Pharmacokinetics

- 1. BAX 855 PK parameters based on FVIII activity at baseline and steady state:
  - AUC0-∞ (Area under the plasma concentration versus time curve from time 0 to infinity), IR (incremental recovery) at 15 30 minutes post-infusion, T<sub>1/2</sub> (plasma half-life), MRT (mean residence time), CL (clearance), maximum plasma concentration (Cmax) and time to maximum concentration in plasma (Tmax), Vss (Volume of distribution at steady state)
  - Incremental recovery (IR) over time

# **8.4.3** Exploratory Outcome Measures

- 1. Thrombin generation assay (TGA) parameters: (lag time, time to peak thrombin generation, peak thrombin generation, and endogenous thrombin potential [ETP])
- 2. Bleed and pain severity scores as measured by the Haemo-SYM questionnaire
- 3. HRQoL as assessed using EQ-5D and mental domain and component scores of SF-36
- 4. Health resource utilization

# 8.5 Randomization and Blinding

This is a randomized, open-label, concurrent, dose regimen comparison clinical study. In order to minimize/avoid bias, once eligibility is confirmed, subjects will be randomly assigned to 1 of 2 treatment regimens with PK-guided dosing targeting FVIII trough levels of 1-3% or approximately 10% (8-12%) in a 1:1 ratio. Randomization occurs after the PK assessment and will be stratified according to subjects' pre-study treatment regimen (prophylaxis vs. on-demand).

# 8.6 Study Stopping Rules

This study will be halted (enrollment and treatment temporarily stopped), pending further review by sponsor, or stopped if the following criterion is met:

- If 2 or more subjects develop a high responder inhibitory antibody > 5 BU, confirmed by 2 measurements within a 2-4 week period at the central laboratory, after BAX 855 administration
- If 2 or more subjects develop anaphylaxis following exposure to BAX 855

The study may be terminated, if 1 or more of the following criteria are met:

- The sponsor decides to terminate the study based upon its assessment of safety
- The sponsor decides to terminate the study for administrative reasons

# 8.7 Investigational Product(s)

# 8.7.1 Packaging, Labeling, and Storage

BAX 855 is formulated as a sterile, highly purified protein preparation in lyophilized form for i.v. infusion and is provided in single-dose vials with a vial of diluent (2 mL or 5 mL SWFI, as available). A butterfly transfer set with luer-lock syringes and a needleless transfer device (BAXJECT II high-flow (HF) or BAXJECT III, as available) will be used for reconstitution and bolus i.v. delivery. The BAXJECT system is a needleless liquid transfer device with the primary function of transferring diluent from its vial into an evacuated vial containing product requiring reconstitution prior to infusion.

A minimum of 4 lots of BAX 855 manufactured for this study will be used. Four potencies of BAX 855 may be used, depending upon availability: 250, 500, 1,000 and 2,000 IU/vial.

The recommended storage conditions for BAX 855 are 2°C to 8°C (36°F to 46°F) and it should not be allowed to freeze. BAX 855 should be stored and protected from light. The reconstituted product should ideally be used immediately but no longer than 3 hours after reconstitution.

For additional information, such as reconstitution instructions, please refer to the BAX 855 IB and/or other specific instructions provided by the sponsor.

#### 8.7.2 Administration

Following reconstitution, BAX 855 should be administered using plastic syringes provided by the sponsor since proteins such as BAX 855 may adhere to the surface of glass syringes. BAX 855 will be administered i.v. using an appropriately sized syringe, as a bolus infusion with a maximum infusion rate of 10 mL/min, as described in the BAX 855 IB. The reconstituted BAX 855 must be administered at room temperature and within 3 hours.

# BAX 855 dose calculation will be based on the stated actual potency of each vial.

# PK assessment and determination of IR

For the PK assessment in individual subjects (initial and at steady state), only vials of the same lot with a nominal potency of 500 IU should preferably be used. If due to a subject's weight, the PK or IR infusion volume will exceed 30 mL, 1000 IU vials should preferably be used to reduce the volume administered.

The total calculated dose may be rounded up or down to the nearest whole vial in case 500 IU potency vials are used. However, in case vials with a nominal potency of 1,000 IU/vial are used, the total calculated dose should not be rounded up or down to the nearest whole vial to ensure accurate dosing (eg, 2.5 vials).

# Infusions for prophylaxis and treatment of bleeding episodes

Two different lots per infusion may be used, however, each vial must be reconstituted with its own kit. The total calculated dose can be rounded up or down to the nearest whole vial.

# 8.7.3 Description of Treatment

Subjects will be randomized to one of two PK-tailored prophylactic dose regimens (see Section 8.5) each of them targeting:

- FVIII trough levels of 1-3% with twice weekly dosing, or
- FVIII trough levels of approximately 10% (8-12%) with dosing every other day.

The individual subject's dose will be calculated by the sponsor and provided to the study site. More frequent dosing should be considered if single doses of 80 IU/kg are required or regular FVIII peak levels of 200 % would be reached or exceeded.

# 8.7.3.1 BAX 855 Dosing for PK Assessment

Following a 72-96 h washout period, depending on the FVIII concentrate, subjects will undergo an initial PK assessment with BAX 855 vi:

At Visit 9 months, ie after 9 months of prophylactic treatment with BAX855, a repeat PK at steady state will be performed. No wash-out period will be required prior to the repeat PK determination; however, the PK infusion should preferably coincide with the prophylactic treatment schedule to ensure that the baseline FVIII trough level is reached.

The BAX 855 dose to be used for the PK assessment is  $60 \pm 5$  IU/kg. It must be administered in the hospital/clinic setting under medical supervision.

# 8.7.3.2 BAX 855 Prophylaxis Dosing

FVIII trough level of 1-3%:

BAX 855 will be administered twice weekly, with either:

- Infusion with alternating 3-days and 4-days infusion intervals; the doses will be different if a 3 or a 4-days interval needs to be covered.
- An infusion every 3.5 days.
- More frequent dosing should be considered if single doses of 80 IU/kg are required or regular FVIII peak levels of 200 % would be reached or exceeded.

#### FVIII trough level of approximately 10% (8% - 12%):

- BAX 855 will be infused every other day.
- A daily dosing may be considered to prevent regular high FVIII peak levels

The required dose and frequency will be provided by the sponsor. Subjects must adhere as closely as possible to the dosing regimen. If a dose is missed, it must be documented and the next dose will be taken as soon as possible. After this dose, the regularly scheduled regimen will be resumed. Subjects requiring treatment for a breakthrough bleeding episode should resume their PK-tailored prophylaxis as soon as the bleeding episode is resolved.

The days of the week on which treatment is administered may be selected by the subject and/or his/her physician and should provide maximum coverage for vigorous activities.

In case a subject underwent a PK determination in any of the BAX855 studies, the PK assessment may have to be repeated based on the sponsor's evaluation.

To provide some flexibility, the weekly schedule in terms of the days of the week may be changed during the course of the study to best accommodate potential changes in the subject's life style. However, the initially calculated and adjusted, if applicable, dose regimen should be maintained.

For each subject, the BAX 855 infusions to perform PKs, IRs and the first individualized prophylaxis dose of BAX 855 at the Baseline visit, which includes an IR assessment, must be administered in the hospital/clinic setting under medical supervision. All other treatments may be self-administered, administered by a parent or caregiver, or administered in the clinic or hospital setting. Each subject's physician will determine the setting of treatment administration. If the subject will self-administer BAX 855, the investigator will ensure that the subject and/or his caregiver have been adequately trained.

The weight determined at screening will be the basis for dose calculation of BAX 855. If there is a  $\pm$  10% change in weight from the screening visit (as measured at a subsequent study visit), the total dose in IU will be recalculated. Similarly, any additional  $\pm$  10% change in weight from this new baseline will result in a dose recalculation.

# 8.7.3.3 BAX 855 Dose and/or Frequency Adjustments

In the first 6-month treatment period the regimen may be adjusted based on the FVIII trough level determined at each study visit. FVIII trough levels should always be determined immediately before the planned next scheduled prophylactic infusion which may coincide with an infusion for determination of IR.

Before dose adjustment, if applicable, a confirmatory FVIII trough level determination at an additional study visit within 2 weeks after receipt of the FVIII activity results has to be performed vii. This additional study visit should also occur after either a 48 h wash-out period in case of an every other day dosing or 72 or 96 hours in case of twice weekly infusions to coincide with the regular prophylactic infusion. After receipt of the repeat FVIII activity results, dose adjustments should be performed:

- If the lower FVIII trough activity level is < 1% and < 8% respectively;
- If the upper FVIII trough activity level exceeds 3% and 12% respectively. Given the assay variations, fluctuations of approximately 3% are possible.

This additional visit may coincide with regular scheduled study visit.

Approximately 2 weeks after the dose adjustment, a repeat FVIII trough level determination at an additional study visit has to be performed, if it does not coincide with the next scheduled study visit. The blood draw for the FVIII trough level measurement should occur after a wash-out period of at least 48 h in case of an every other day dosing or 72 or 96 hours in case of twice weekly infusions to coincide with the regular prophylactic infusion.

Dose adjustments in the second 6-month period may only be performed if FVIII trough levels are considerably below the required FVIII trough levels of 1% and 8%. Should the upper limit considerably exceed 3% and 12% respectively, a dose adjustment may be performed.

In case, the FVIII levels are below the required lower limit, the BAX 855 dosage may be increased up to a maximum of  $80 \pm 5$  IU/kg and/or the dosing frequency may be increased. Doses as high as 80 IU/kg may be used, provided the FVIII peak level does not exceed 200%. Otherwise, the frequency of prophylactic infusions has to be increased.

A detailed procedure for dose adjustment will be provided in a separate document.

In subjects with severe hemophilic arthropathy and/or target joints viii who continue to experience recurrent bleeding episodes, an imaging technology such as MRI or ultrasound of the affected joint(s) has be applied to verify the presence of a bleed.

Also, if at any time during the course of the study, a subject's starts to experience an unexpected high bleeding rate or experience bleeding episodes that do not adequately respond to BAX855 therapy, he/she will be evaluated for the presence of inhibitory and total binding antibodies to FVIII, BAX855 and PEG, and clinically managed at the discretion of the investigator. It is also recommended to perform an incremental recovery.

# 8.7.3.4 Treatment of Bleeding Episodes

BAX 855 ( $10-60 \pm 5$  IU/kg) will be used for treatment of bleeding episodes (ie, breakthrough bleeding episodes during prophylaxis) according to the guidelines in Table 1. These guidelines may be adjusted by the investigator based upon his or her clinical judgment.

It is critical that treatment of a bleed is initiated as soon as possible after occurrence of the bleeding episode.

viii A target joint is defined as a single joint (ankles, knees, hips, or elbows) with ≥ 4 spontaneous bleeding episodes in any consecutive 6-month period.
When bleeding is controlled, additional infusions of BAX 855 to maintain hemostasis are permitted, if required. Infusions given to maintain hemostasis should be documented in the eCRF.

For a detailed description of bleeding episodes into different sites see Supplement 22.

| Table 1 BAX 855 Treatment Guidelines for Bleeding Episodes | | |
|---|---|---|
| Type of Bleeding Episode | FVIII Level Required (%) Dose (IU/kg) | Frequency of Dosing |
| Minor Early hemarthrosis, mild muscle bleeding, or mild oral bleeding, including, epistaxis | 20 to 40% 10 to 20 (±5) IU/kg | Repeat infusions every 12 to 24 h for 1 to 3 days until the bleeding episode is resolved |
| Moderate Moderate bleeding into muscles, bleeding into the oral cavity, definite hemarthrosis, and known trauma | 30 to 60%<br>15 to 30 (±5) IU/kg | Repeat infusions every 12 to 24 h for 3 days or more until the pain and acute disability/incapacity are resolved |
| Major Significant gastrointestinal bleeding, intracranial, intra-abdominal, or intrathoracic bleeding, central nervous system bleeding, bleeding in the retropharyngeal or retroperitoneal spaces or iliopsoas sheath, fractures, head trauma | 60 to 100% 30 to 60 (±5) IU/kg In case of life-threatening bleeds, a dose of 80 (±5) IU/kg may be considered | Repeat infusions every 8 to 12 h until the bleeding episode/threat is resolved |

The required units will be calculated according to the following formula:

body weight (kg) x desired FVIII rise (%) (IU/dL) x {reciprocal of observed recovery}

Whenever possible, the subject's most recent individual IR should be used. In its absence, an anticipated recovery of 2.5 (IU/dL)/(IU/kg) based on the initial PK with BAX855 in the Phase 2/3 pivotal study, should be assumed and the required units calculated using the following formula:

body weight (kg) x desired FVIII rise (%or (IU/dL) x 0.4 dL/kg

The amount to be administered and the frequency of administration should always be oriented to the clinical effectiveness in the individual case.

In subjects with severe hemophilic arthropathy and/or target joints with recurrent bleeding requiring more than 2 infusions per bleed and/or where efficacy ratings are generally fair or none, an imaging technology such as MRI or an ultrasound of the affected joint(s) has to be applied to verify the presence of a bleed.

## 8.7.3.5 Treatment for Surgery or Dental Procedures

Subjects enrolled into this BAX 855 study (261303) and who require planned surgery or dental procedures will be treated according to the treatment recommendations including a FVIII substitution plan described in Supplement 22.

## 8.7.3.6 Immune Tolerance Induction for Inhibitor Development.

Subjects who develop a confirmed (ie, 2 separate assessments within a 2 to 4 week period from the central laboratory) high responder inhibitor (>5 BU) or low responder inhibitor ( $\le5$  BU but  $\ge0.6$  BU) that cannot be adequately managed by the protocol-required prophylactic regimen with BAX 855 will be discontinued from this study. The decision to initiate immune tolerance induction (ITI) with ADVATE will be made by the subject's physician, and may be discussed with the sponsor's medical director prior to initiation. The regimen used for ITI will be determined by the treating physician but should be discussed with the sponsor's medical director. ITI is not within the scope of this study.

## **8.7.4** Investigational Product Accountability

The investigator will ensure that the IP (BAX 855) is stored as specified in the protocol and that the storage area is secured, with access limited to authorized study personnel. The investigator will maintain records that the IP was received, including the date received, drug identity code, date of manufacture or expiration date, amount received and disposition. IP must be dispensed only at the study site or other suitable location (eg, infusion center; home, as applicable per study design). Records will be maintained that includes the subject identification code (SIC), dispensation date, and amount dispensed. All remaining partially used and/or unused IP will be returned to the sponsor or sponsor's representative after study completion/termination, or destroyed with the permission of the sponsor in accordance with applicable laws and study site procedures. If IP is to be destroyed, the investigator will provide documentation in accordance with sponsor's specifications.

#### 8.8 Source Data

Per ICH GCP, source data are defined as all information in original records and certified copies of original records of clinical findings, observations, or other activities in a clinical trial that are necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents (original records or certified copies), which may be in paper and/or electronic format. Source data for this study comprise the following: hospital records, medical records, clinical and office charts, laboratory notes, memoranda, subjects' diaries or evaluation checklists, outcomes reported by subjects, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate copies, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files, and records kept at the pharmacy, at the laboratories and at medico-technical departments involved in the clinical study.

For additional information on study documentation and CRFs, see Section 18.2. The use of subject diaries is described in Section 10.5.

## 9. SUBJECT SELECTION, WITHDRAWAL, AND DISCONTINUATION

#### 9.1 Inclusion Criteria

## 9.1.1 Subjects Transitioning from Another BAX 855 Study

Subjects transitioning from another BAX 855 study who meet **ALL** of the following criteria are eligible for this study:

- 1. Subject has completed the end of study visit of a BAX 855 study or is transitioning from the ongoing Baxalta Continuation Study 261302.
- 2. Subject is either receiving on-demand treatment or prophylactic treatment with BAX 855 and had an ABR of  $\geq 2$  documented and treated during the past 12 months.
- 3. Subject is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count  $\geq$  200 cells/mm<sup>3</sup>, as confirmed by central laboratory.
- 4. Subject is willing and able to comply with the requirements of the protocol.

# 9.1.2 Inclusion Criteria for Newly Recruited Subjects

Newly recruited subjects including BAX855 naïve subjects who meet **ALL** of the following criteria are eligible for this study:

- 1. Subject is 12 to 65 years old at the time of screening
- 2. Subject has severe hemophilia A (FVIII clotting activity < 1%) as confirmed by central laboratory or by historically documented FVIII clotting activity performed by a certified clinical laboratory and/or a FVIII gene mutation consistent with severe hemophilia A
- 3. Subject has been previously treated with plasma-derived FVIII concentrates or recombinant FVIII for ≥ 150 documented exposure days (EDs)
- 4. Subject is either receiving on-demand treatment or prophylactic treatment and had an annual bleeding rate of  $\geq 2$  documented and treated during the past 12 months.
- 5. Subject has a Karnofsky performance score of  $\geq$  60 at screening
- 6. Subject is HIV-; or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm3, as confirmed by central laboratory at screening
- 7. Subject is hepatitis C virus negative (HCV-) by antibody (if positive, additional PCR testing will be performed), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis
- 8. If female of childbearing potential, subject presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study
- 9. Subject is willing and able to comply with the requirements of the protocol.

#### 9.2 Exclusion Criteria

# 9.2.1 Exclusion Criteria for Subjects Transitioning from Another BAX 855 Study

Subjects transitioning from another BAX 855 study who meet **ANY** of the following criteria are not eligible for this study:

- 1. Subject has developed a confirmed inhibitory antibody to FVIII with a titer of ≥ 0.6 BU using the Nijmegen modification of the Bethesda assay as determined at the central laboratory during the course of the previous BAX 855 study.
- 2. Subject has been diagnosed with an acquired hemostatic defect other than hemophilia A.
- 3. The subject's weight is < 35 kg or > 100 kg.
- 4. Subject's platelet count is < 100,000/mL.
- 5. Subject has an abnormal renal function (serum creatinine > 1.5 times the upper limit of normal).
- 6. Subject has active hepatic disease with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels  $\geq 5$  times the upper limit of normal.
- 7. Subject is scheduled to receive a systemic immunomodulating drug (e.g. corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or α-interferon) other than anti-retroviral chemotherapy during the study.
- 8. Subject has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject's safety or compliance.
- 9. Subject is planning to take part in any other clinical study during the course of the study.
- 10. Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

## 9.2.2 Exclusion Criteria for Newly Recruited Subjects

Newly recruited subjects who meet **ANY** of the following criteria are not eligible for this study:

1. Subject has detectable FVIII inhibitory antibodies (≥ 0.6 BU using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening.

- 2. Subject has a history of confirmed FVIII inhibitors with a titer ≥ 0.6 Bethesda Units (BU) (as determined by the Nijmegen modification of the Bethesda assay or the assay employed with the respective cut-off in the local laboratory) at any time prior to screening.
- 3. Subject has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease).
- 4. The subject's weight is < 35 kg or > 100 kg.
- 5. Subject's platelet count is < 100,000/mL.
- 6. Subject has known hypersensitivity towards mouse or hamster proteins, PEG or Tween 80.
- 7. Subject has severe chronic hepatic dysfunction [eg,  $\geq$  5 times upper limit of normal alanine aminotransferase (ALT) or aspartate aminotransferase (AST), as confirmed by central laboratory at screening, or a documented INR > 1.5].
- 8. Subject has severe renal impairment (serum creatinine > 1.5 times the upper limit of normal).
- 9. Subject has current or recent (< 30 days) use of other pegylated drugs prior to study participation or is scheduled to use such drugs during study participation.
- 10. Subject is scheduled to receive during the course of the study, a systemic immunomodulating drug (e.g. corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day, or  $\alpha$ -interferon) other than anti-retroviral chemotherapy.
- 11. Subject has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
- 12. Subject has a medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance.
- 13. Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

#### 9.3 Withdrawal and Discontinuation

Any subject may voluntarily withdraw (ie, reduce the degree of participation in the study) consent for continued participation and data collection. The reason for withdrawal will be recorded on the End of Study CRF. Assessments to be performed at the termination visit (including in cases of withdrawal or discontinuation) are described in Section 10.6 and Section 21.3.

Discontinuation (ie, complete withdrawal from study participation) may be due to dropout (ie, active discontinuation by subject) or loss to follow-up (ie, discontinuation by subject without notice or action). Additionally, the investigator and sponsor have the discretion to discontinue any subject from the study if, in their judgment, continued participation would pose an unacceptable risk for the subject.

Subjects also will be withdrawn from treatment or discontinued from further study participation for the following reasons:

- The subject develops a confirmed high responder inhibitory antibody to FVIII (> 5 BU by Nijmegen modification of the Bethesda assay) or a low responder inhibitory antibody (≤ 5 BU but ≥ 0.6 BU) that cannot be managed by the protocol-required prophylactic dosing.
- The subject experiences a severe anaphylactic reaction to BAX 855.
- The subject requires therapy with another pegylated product (eg, PEG-Interferon).
- The subject frequently misses administration of IP (misses more than 30% of planned prophylactic doses within any 3-month period).
- The subject is non-compliant with study procedures, in the opinion of the investigator and/or sponsor.
- The subject uses his/her usual FVIII therapy following the baseline infusion
- The subject requires major emergency surgery during this study
- The subject experiences a life-threatening bleeding episode (eg, any gastrointestinal hemorrhage or intracranial hemorrhage) requiring the use of a FVIII concentrate other than BAX855.
- The subject experiences severe trauma requiring extensive FVIII replacement therapy other than BAX855

#### 10. STUDY PROCEDURES

#### 10.1 Informed Consent and Enrollment

Any patient, or their legal representatives, as required, who provides informed consent (ie, signs and dates the informed consent form and assent form, if applicable) is considered enrolled in the study.

# 10.2 Subject Identification Code

The following series of numbers will comprise the SIC: protocol identifier (ie, 261303) to be provided by the sponsor, 3-digit number study site number (eg, 002) to be provided by the sponsor, and 3-digit subject number (eg, 003) reflecting the order of enrollment (ie, signing the informed consent form). For example, the third subject who signed an informed consent form at study site 02 will be identified as Subject 261303-002003. All study documents (eg, CRFs, clinical documentation, sample containers, drug accountability logs, etc.) will be identified with the SIC. Additionally, a uniquely coded SIC(s) is permitted as long as it does not contain a combination of information that allows identification of a subject (eg, collection of a subject's initials and birth date would not be permitted), in compliance with laws governing data privacy.

## 10.3 Screening and Study Visits

The study site is responsible for maintaining an enrollment/screening log that includes all subjects enrolled. The log also will serve to document the reason for screening failure. If a subject does not satisfy all screening criteria, the same subject may be re-screened at a later date. A complete or partial re-screen may also become necessary at the discretion of the investigator or sponsor. All screening data will be collected and reported in eCRFs, regardless of screening outcome. For the purpose of analysis, only the data from the most recent screening visit will be used. If a subject is re-screened, the End of Study CRF should be completed, and a new ICF, new SIC and new CRF are required for that subject.

The screening procedures including laboratory evaluations must be completed within 56 days or repeated if more than 56 days have elapsed. Exemptions may be granted for administrative reasons, eg, delay in timely availability of laboratory results.

The overall study design is illustrated in the Figure 1. Details on the procedures to be performed at each study visit, including screening, can be found in Supplement 21.2 Detailed Flow Diagram of Study Procedures, Supplement 21.3 Schedule of Study Procedures and Assessments, and Supplement 21.4 Clinical Laboratory Assessments. Only explanatory details are provided in the section below.

# 10.3.1 Subjects Transitioning from Other BAX 855 Studies

Subjects transitioning from other BAX 855 studies ix can use the end of study assessments in their previous BAX 855 study for screening visit assessments in this PK-guided study. Any additionally required screening assessments will be performed the same day. Subjects will return to the study site no later than 56 days for the conductance of the PK assessment, if applicable, provided eligibility has been confirmed. At the screening visit the subject will be supplied with study IP of study 261303. Until the baseline visit subjects will be treated according to their previous BAX 855 treatment regimen.

## **10.3.2** Newly Recruited Subjects

Newly recruited subjects will continue using their FVIII treatment regimen until baseline/start of PK guided prophylaxis, except for one infusion with BAX 855 for PK determination.

## **10.4 Medications and Non-Drug Therapies**

The following medications and non-drug therapies are **not** permitted within 30 days before study entry and during the course of the study:

- Medications:
  - ➤ Any pegylated medication (eg, PEG-interferon) except BAX 855 for transitioning subjects
  - ➤ Any investigational drug, biologic, or device except BAX 855 for transitioning subjects

A subject who has taken any of these medications or received any of these non-drug therapies will be considered a protocol deviation.

The use of any FVIII concentrate other than BAX 855 during the course of the study following the first BAX 855 PK guided prophylactic infusion at baseline will result in the immediate withdrawal of the subject. Every effort should be made to have the Completion/Termination Visit performed. The use of (commercial) ADVATE may be permitted for a short period of time for administrative reasons.

The following medications and non-drug therapies are permitted before study entry and during the course of the study:

Medications:

For subjects in the continuation study, data from a regular scheduled study visit can be used as long they are not older than 4 weeks prior to screening.

- ➤ Hemostatic agents, such as tranexamic acid, are permitted, as indicated by the subject's treating physician, to treat mucosal bleeding or during perioperative management during the study
- Any medications deemed necessary by the subject's physician to treat or prevent any medical condition
- Any over-the-counter medication used by the subject to treat symptoms or signs
- > Supplemental vitamins, minerals
- Non-drug therapies:
  - Any non-drug therapy (eg, physiotherapy) deemed necessary by the subject's physician to treat or prevent any medical condition

# 10.5 Subject Diary and Patient Reported Outcomes

A subject diary will be provided to each subject at the Screening Visit to record the following information:

- 1. Infusion record for BAX 855
- 2. Details of bleeding episodes and response to treatment. For a detailed description of bleeding episodes into different sites see Supplement 22.
- 3. Physical activity within 8 h prior to the occurrence of a bleeding episode
- 4. Untoward events
- 5. PROs (see Section 10.5.1)

For each bleeding episode, the following information will be recorded by the subject/subject's caregiver or by authorized, qualified personnel at the study site:

- Location of bleed, eg, joint, soft tissue, muscle, body cavity, intracranial, other.
- Type of bleed, ie, spontaneous (i.e. not related to injury/trauma), injury (definitely due to injury/trauma).
- Severity of bleed, eg, minor, moderate, major (see Table 1).
- Date and time of onset of bleed.
- Date and time of each infusion of BAX 855 required to achieve adequate hemostasis.
- Date and time of resolution of bleeding episode.
- Overall clinical efficacy rating according to the rating scale as described in Table 2 at 24 (±2) hours after initiation of treatment and at resolution of bleed.
- Physical activity within 8 h prior to the occurrence of the bleeding episodes.

Subjects and/or their legally authorized representatives will be trained on use of the diary. The diary will be provided in electronic or paper format and remain with the subject for the duration of the study. The investigator will review the diary for completeness and request missing information periodically and in a timely manner. Untoward events recorded in the diary will be reported as AEs according to the investigator's discretion and clinical judgment. Subject entries in the diary will serve as source records. If ediaries are used, during study participation the investigator has access to the database holding the subject diary data. After study closure, the investigator will receive the diary records for their subjects, including audit trail records, in PDF format. The data will be transmitted to the CRF by a validated transfer.

## **10.5.1 Patient Reported Outcomes**

The PRO instruments to be measured in this study are described below. These measures will be administered in this study at 3 time points: Screening or Baseline Visit, 6-month visit, and Completion/Termination Visit, whereas the EQ-5D, Patient Activity Level, and Health Resource Use will be measured prior at each study visit before study specific procedures are started. Note that due to the unavailability of linguistically validated translations of certain PRO measures in certain countries, some of these questionnaires may not be administered in all countries participating in this study. In addition, subjects who are younger than the minimal age limit required for these assessments will not be required to complete the assessment.

- Haemo-SYM Questionnaire This is a self-administered, validated questionnaire designed to assess symptom severity in patients with hemophilia. This measure contains 17 items and includes 2 domains: Bleeds and Pain. Scores for each of these 2 domains can be calculated, with higher scores indicating more severe symptoms. This questionnaire will be administered only to subjects ≥18 years of age.
- 2. **Short Form-36 (SF-36)** The SF-36 is a self-administered, validated questionnaire designed to measure generic HRQoL. This 36-item questionnaire measures 8 domains, including: Physical functioning, Role-physical, Bodily pain, General health, Vitality, Social functioning, Role emotional, and Mental health. Two summary scores can be calculated, the Physical Component Score, and the Mental Component Score. Additionally, scores can be calculated for each of the 8 domains. Higher scores indicate better health status. This questionnaire will be administered only to subjects ≥14 years of age.

3. **EQ-5D Questionnaire** – The EQ-5D is a self-administered, standardized measure of health status that provides a generic measure of health for clinical and economic appraisal consisting of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression each with 5 levels. There is an additional EQ VAS to record how good or bad their health state is.

## 4. Patient Activity Level

Subjects will also be asked to estimate their activity levels. This will consist of a few questions asking subjects to rate their current level of activity. These data will be collected for all age groups.

5. **Health Resource Use** – For each occurrence (throughout the study), the subject will record the following events: days missed from work/school (as appropriate) and days not able to perform normal activities outside of work/school due to hemophilia, physician office visits, hemophilia treatment site visits, emergency room visits (reason and number), and hospitalizations (reason, dates of hospitalization and associated length of stay).

## **10.6 Subject Completion/Discontinuation**

A subject is considered to have completed the study when he/she ceases active participation in the study because the subject has, or is presumed to have, completed all study procedures according with the protocol (with or without protocol deviations).

Reasons for completion/discontinuation will be reported on the Completion/Discontinuation CRF, including: completed, screen failure, AE (eg, death), discontinuation by subject (eg, lost to follow-up [defined as 3 documented unsuccessful attempts to contact the subject], dropout), physician decision (eg, pregnancy, progressive disease, non-compliance with IP/protocol violation(s), recovery), study terminated by sponsor, or other (reason to be specified by the investigator, eg, technical problems). Regardless of the reason, all data available for the subject up to the time of completion/discontinuation should be recorded on the appropriate eCRF.

Every effort will be made to have discontinued subjects complete the study completion/termination visit. If the completion/termination visit is done as an additional, unscheduled visit, the assessment results shall be recorded with the completion/termination visit. If a subject terminates participation in the study and does not return for the completion/termination visit, their last recorded assessments shall remain recorded with their last visit. The reason for discontinuation will be recorded, and the data collected up to the time of discontinuation will be used in the analysis and included in the clinical study report.

If additional assessments are required, the assessments shall be recorded separately. Assessments to be performed at the termination visit (including in cases of withdraw or discontinuation) can be found in Supplement 21.2 Detailed Flow Diagram of Study Procedures, Supplement 21.3 Schedule of Study Procedures and Assessments, and Supplement 21.4 Clinical Laboratory Assessments.

In the event of subject discontinuation due to an AE, clinical and/or laboratory investigations that are beyond the scope of the required study observations/assessments may be performed as part of the evaluation of the event. These investigations will take place under the direction of the investigator in consultation with the sponsor, and the details of the outcome may be reported to the appropriate regulatory authorities by the sponsor.

## 10.7 Procedures for Monitoring Subject Compliance

Subject compliance with the BAX 855 individualized treatment regimens will be monitored by review of subject diaries and by IP accountability.

#### 11. ASSESSMENT OF EFFICACY

# 11.1 Bleeding Assessment

Each individual bleed, spontaneous or traumatic, will be recorded in the subject's diary, and/or recorded in physician/nurse/clinic notes. A bleed is defined as subjective (eg, pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII. For further definitions of bleeds see Supplement 22. Bleeds occurring at the same anatomical location (eg, right knee) with the same etiology (ie, spontaneous vs. injury) within 72 h of onset of the first bleed will be considered a single bleed.<sup>31</sup> A new bleed is defined as a bleed occurring > 72 hours after stopping treatment for the original bleed for which treatment was initiated and had an initial moderate to excellent response to treatment.<sup>31</sup> Bleeding occurring at multiple locations related to the same injury (eg, knee and ankle bleeds following a fall) will be counted as a single bleeding episode.

The subject will also indicate in the diary on a preselected scale the type of activity within 8 hours prior to the bleeding episode.

For the primary assessment, the total bleed rate in the second 6-month study period will be calculated (ie, after the 6-month visit to the Completion/Termination Visit). The secondary outcome measures, spontaneous and traumatic ABR, and spontaneous AJBR will also be calculated from the recorded bleeds.

## 11.1.1 Hemostatic Efficacy Rating for Treatment of Bleeding Episodes

The subject or their caregiver will rate the severity (minor, moderate, or major) of the bleeding episode and will rate the overall treatment response at  $24 (\pm 2)$  hours after the initiation of treatment and at the resolution of bleed using a 4-point efficacy rating scale (Table 2). Since the efficacy rating is based to a large degree on cessation of pain, the investigator/subject shall, in particular in case of injury-related bleeding into one or more than one location, consider the injury-related symptoms when performing the efficacy rating 24 hours after initiating treatment and at resolution of bleed.

As per Table 2, multiple infusions of BAX 855 may be administered for the treatment of a bleeding episode. The overall response to all infusions combined is the rating that will be recorded at resolution of bleed.

| Table 2 Efficacy Rating Scale for Treatment of Bleeding Episodes | |
|---|---|
| Excellent | Full relief of pain and/or cessation of objective signs of bleeding (eg, swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage) after a single infusion. No additional infusion is required for the control of bleeding. Administration of further infusions to maintain hemostasis would not affect this scoring. |
| Good | Definite pain relief and/or improvement in signs of bleeding after a single infusion. Possibly requires more than 1 infusion for complete resolution. |
| Fair | Probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion. Required more than 1 infusion for complete resolution. |
| None | No improvement or condition worsens. |

Details pertaining to all treatments for each bleed, including response to treatment, will be recorded by study subjects/subjects' caregiver in subject diaries provided by the sponsor or sponsor's representative. At each study visit, the investigator will review together with the subject/subject's caregiver the response to treatment and evaluate the hemostatic efficacy rating. It may become necessary to re-discuss the rating with the subject/subject's caregiver to ensure the Rating Scale is fully understood:

- Any inconsistency between the efficacy rating and the number of infusions used to treat a bleeding episode, or a response to treatment rated as "none" must be immediately clarified.
- If 2 or more responses to treatment of unique bleeding episodes are rated "fair", the investigator may re-evaluate the dosing regimen and the time from bleeding onset to the start of treatment. If a bleeding episode requires only one infusion but response to treatment is rated "fair", the rating should be evaluated and the Rating Scale should be reviewed with the subject/subject's caregiver.

If more than one infusion was given to treat a bleeding episode, and the treatment was rated "excellent", additional information should be provided about the severity of the bleeding episode (see Table 1) and/or whether additional infusions were given to maintain hemostasis. If infusions were given to maintain hemostasis after resolution of bleed, this should be recorded accordingly in the eCRF.

# 11.1.2 Number of BAX 855 Infusions Needed for the Treatment of Bleeding Episodes

The number of BAX 855 infusions needed for each bleeding episode depends on the severity and location of the bleed and is determined by the subject, his/her caregiver, and/or clinician treating the subject, and is based upon the subject's response to treatment, using the Efficacy Rating Scale for Treatment of Bleeding Episodes in Table 2. An infusion is defined as completion of administration of the calculated dose of BAX 855. If an infusion is interrupted, eg, due to vascular access issues, and must be restarted, it will be recorded as 1 infusion. If an infusion is terminated for any reason prior to completion of infusion and not restarted, it will be recorded as an infusion; reasons for not completing the infusion will be recorded.

# 11.1.3 Hemophilia Joint Health Score (HJHS)

The HJHS will be assessed at Baseline, ie the first PK guided prophylactic infusion with BAX855, and the completion/termination visit. An X-ray of an impaired joint will be taken for assessment of joint status. In addition, the PI or a qualified staff member (e.g. physiotherapist) will assess the following components of the elbow, knee, and ankle joints: swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain, and strength, together with an assessment of the global gait.

## 11.1.4 Weight-Adjusted Consumption of BAX 855

Weight-adjusted consumption of BAX 855 will be determined based upon the record in subjects' diaries of the amount of BAX 855 infused and the subject's weight, as measured in the clinic.

#### 11.1.5 Peri-operative efficacy assessments

For the detailed description of intra-, post- and perioperative efficacy see Supplement 22.

# 12. DETERMINATION OF FVIII AND VWF ANTIGEN, FVIII ACTIVITY AND TGA

#### 12.1 PHARMACOKINETICS

An initial evaluation of PK parameters based on FVIII activity will be performed in all subjects prior to randomization<sup>x</sup>. This PK will be performed following a wash-out period of at least 72-96 hours, depending on the type of FVIII concentrate used.

In all subjects, a repeat PK evaluation will be performed at the 9 month  $\pm$  2 weeks visit to assess PK at steady state. For the repeat PK no wash-out period will be required and the PK infusion should coincide with the scheduled prophylactic infusion to ensure that the trough FVIII activity level is determined, eg 2 days following the most recent infusion in the intensified treatment group with targeted FVIII trough levels between 8-12%.

Samples will be taken to assess FVIII activity, FVIII antigen and TGA parameters preinfusion and at several time points post-infusion over a 4-day period following a single dose of  $60 \pm 5$  IU/kg of BAX 855. VWF antigen will be also determined from the preinfusion blood sample.

Blood samples are collected at the following time points:

| Table 3 PK Time Points | | | | |
|---|---|---|---|---|
| | | FVIII (Activity and Antigen) | VWF Antigen | TGA |
| Pre-infusion | Within 30 minutes prior to infusio | + | + | + |
| Infusion | 60±5 IU/kg of BAX855 | | | |
| Post-infusion | 15 – 30 minutes | + | | + |
| | 3 hours $\pm$ 30 minutes | + | | + |
| | 8 hours ± 30 minutes | + | | + |
| | 24 hours ± 2 hour | + | | + |
| | 48 hours ± 4 hour | + | | + |
| | 72 hours ± 4 hour | + | | + |
| | 96 hours ± 4 hour | + | | + |

In case a subject underwent a PK determination in BAX855 surgery or continuation study, the PK assessment may have to be repeated based on the sponsor's evaluation.

The PK infusion may be administered via a central line or a peripheral vein. Upon completion of the infusion, the butterfly catheter should be flushed with at least 2 mL of saline solution. All PK samples will be collected through a peripheral vein. Blood samples drawn during the first 3 hours after BAX 855 administration will be drawn from a peripheral vein in an extremity distinct from the one that was used for product infusion. After that time, a vein in any appropriate extremity may be used. In the event that a blood sample must be drawn through the central or peripheral line used for administration of IP, the line must first be flushed with 5 mL normal saline or other suitable catheter flush solution that does not contain anticoagulant. At least 5 mL of whole blood must be collected and discarded prior to obtaining the blood sample.

For further details regarding analysis of FVIII activity see Section 13.9.5.

Subjects who have a bleeding episode during the PK assessment period will not have subsequent PK blood samples taken. They will be treated for the bleeding episode, as appropriate (ie, for subjects that transitioned from a previous BAX 855 study, the bleed will be treated with BAX 855; for newly recruited subjects, the bleed will be treated with their current FVIII concentrate). Subsequently, once recovered, subjects will be reinfused for PK assessment following a washout period of at least 84 to preferably 96 hours following the previous dose of BAX 855 or at least 72 hours following the previous dose of another FVIII concentrate. However, depending on the time point of the bleeding episode during the PK evaluation, an exemption may be granted by the sponsor.

#### 12.2 Incremental Recovery (IR)

IR will be determined at each study visit except study visit week  $4\pm 5$  days, week  $8\pm 1$ , and month 4.5 months  $\pm 2$  weeks when only trough levels will be measured. Following a wash-out period required for the respective treatment group, blood samples for the determination of IR will be taken at the following time points:

| Table 4 IR Time Points | | | | |
|---|---|---|---|---|
| | | FVIII (Activity and Antigen) | VWF Antigen | TGA |
| Pre-infusion | Within 30 minutes prior to infusion | + | + | + |
| Infusion | 60±5 IU/kg of BAX855 | | | |
| Post-infusion | 15 -30 minutes | + | | + |

# 12.3 Trough Levels

At study visit week  $4\pm5$  days, week  $8\pm1$  and month  $4.5\pm2$  weeks, FVIII activity trough levels will be measured to ensure that FVIII trough levels are within their targeted range. The blood sampling for FVIII activity, TGA parameters and VWF antigen should be performed immediately prior to the next regular prophylactic infusion, thus maintaining the treatment regimen-specific interval defined for each subject. Following dose adjustments, a FVIII trough level has to be determined approximately 2 weeks following the dose adjustment.

Details on the sampling of blood for determination of FVIII trough levels are presented in Supplement 21.3 and Supplement 21.4

#### 13. ASSESSMENT OF SAFETY INCLUDING IMMUNOGENICITY

# 13.1 Immunogenicity

Immunogenicity of BAX 855 will be assessed prior to the infusion of BAX855 following a washout period of at least 48 h (at steady state in case of every other day dosing) or 72-96 hours (in case of twice weekly infusions) by measurement of the following antibodies (see also Section 21.4 for the time points):

- Inhibitory antibodies to FVIII –using the Nijmegen modification of the Bethesda assay
- Binding antibodies to FVIII, BAX 855, and PEG. Both IgG and IgM antibodies will be measured using an ELISA assay
- Anti-CHO antibodies measured by an ELISA assay

In addition to the time points as described in Section 21.4, the subject should be evaluated for inhibitory and binding antibodies to FVIII, BAX855 and PEG if clinically indicated, eg lack of response to treatment.

A low titer (responder) inhibitor is defined as  $\geq 0.6$  BU but  $\leq 5$  BU. A high titer (responder) inhibitor is defined as  $\geq 5$  BU by Nijmegen modification of the Bethesda assay. Inhibitors must be documented at 2 separate time points within a 2 to 4 week period at a central laboratory. Every confirmed FVIII inhibitor  $\geq 0.6$  BU must be reported as an SAE.

Based on the variability of the binding antibody tests, only samples with titers  $\geq 1:80$  can be confirmed and will be evaluated as positive. IgG subclass 1-4, IgA (using ELISA) and IgE antibodies (using ImmunoCaps, Thermo Fisher) may be assayed as clinically indicated.

The assay for antibodies to CHO protein will use CHO protein derived from cultures of untransfected cells. Testing for binding of anti-CHO protein antibodies will be performed on citrate-anti-coagulated plasma using an ELISA employing polyclonal anti-human IgG antibodies. Antibody-containing samples will be identified in a screening assay followed by a confirmatory assay to exclude false positive results.

All assays will be performed in a central laboratory.

#### 13.2 Adverse Events

#### 13.2.1 Definitions

An AE is defined as any untoward medical occurrence in a subject administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP.

#### 13.2.1.1 Serious Adverse Event

A **serious** adverse event (SAE) is defined as an untoward medical occurrence that at any dose meets one or more of the following criteria:

- Outcome is fatal/results in death (including fetal death)
- Is life-threatening defined as an event in which the subject was, in the judgment of the investigator, at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death had it been more severe.
- Requires inpatient hospitalization or results in prolongation of an existing hospitalization inpatient hospitalization refers to any inpatient admission, regardless of length of stay.
- Results in persistent or significant disability/incapacity (ie, a substantial disruption of a person's ability to conduct normal life functions)
- Is a congenital anomaly/birth defect
- Is a medically important event a medical event that may not be immediately life-threatening or result in death or require hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the definitions above. Examples of such events are:
  - ➤ Intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependence or drug abuse
  - ➤ Reviewed and confirmed seroconversion for human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), hepatitis E virus (HEV), or parvovirus B19 (B19V)
  - $\triangleright$  Development of a confirmed inhibitor to FVIII with an inhibitor level  $\ge 0.6$  BU, as measured by the Nijmegen modification of the Bethesda assay
  - ➤ Severe hypersensitivity/allergic reactions to BAX 855

Uncomplicated pregnancies, following maternal exposure to IP are not considered an (S)AE; however, any pregnancy complication or pregnancy termination by therapeutic, elective, or spontaneous abortion shall be considered an SAE.

#### 13.2.1.2 Non-Serious Adverse Event

A **non-serious** AE is an AE that does not meet the criteria of an SAE.

## 13.2.1.3 Unexpected Adverse Events

An unexpected adverse event is an AE whose nature, severity, specificity, or outcome is not consistent with the term, representation, or description used in the Reference Safety Information (eg, IB, package insert). "Unexpected" also refers to the AEs that are mentioned in the IB as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

For the purposes of this study, all AEs including unexpected AEs experienced by a subject undergoing study treatment will be recorded on the AE CRF.

## 13.2.1.4 Preexisting Diseases

Preexisting diseases that are present before entry in to the study are described in the medical history, and those that manifest with the same severity, frequency, or duration after IP exposure, will not be recorded as AEs. However, when there is an increase in the severity, duration, or frequency of a preexisting disease, the event must be described on the AE CRF.

#### 13.2.2 Assessment of Adverse Events

For the purposes of this study, the following non-serious events experienced after the first IP exposure will not be considered AEs, and thus, not included in the analysis of AEs:

- Hospital or clinic visits for administration of BAX 855
- Hospitalization for routine bleeding episode management that could be managed in the clinic or home-setting but for which the subject was hospitalized
- Hospitalizations for planned medical or surgical procedures, eg, placement of a central venous line (however, when there is an increase in the severity, duration, or frequency of a preexisting disease, the event must be described on the AE CRF)
- Hospitalization or prolongation of hospitalization intended only for social reasons.

- Seroconversion after documented HAV/HBV vaccination prior to or during the study period
- Bleeding episodes/hemophilia-related events: Bleeding episodes are part of the underlying disease and therefore are not AEs. If a bleeding episode was caused by an injury (eg, a fall), the injury would not be reported as an AE, unless it resulted in a medical finding other than a bleeding episode (eg, abrasion of skin; fractured tibia). Therefore, any hemophilia-related event (eg, hemarthrosis, bruising, hemorrhage) will not be reported as an AE, but these events will be recorded on the bleeding event CRF. However, hemophilia-related events meeting the criteria for seriousness (eg, a gastrointestinal hemorrhage requiring hospitalization) will be reported as SAEs and described on the SAE report

All other AEs from the first IP exposure until study completion/discontinuation will be described on the AE CRF using the medical diagnosis (preferred), or, if no diagnosis could be established at the time of reporting the AE, a symptom or sign, in standard medical terminology in order to avoid the use of vague, ambiguous, or colloquial expressions (see definition in Section 13.2). Each AE will be evaluated by the investigator for:

- Seriousness as defined in Section 13.2.1.1
- Severity as defined in Section 13.2.2.1
- Causal relationship to IP exposure or study procedure as defined in Section 13.2.2.2

For each AE, the outcome (ie, recovering/resolving, recovered/resolved, recovered/resolved with sequelae, not recovered/not resolved, fatal, unknown) and if applicable action taken (ie, dose increased, dose not changed, dose reduced, drug interrupted, drug withdrawn, not applicable, or unknown) will also be recorded on the AE CRF. Recovering/resolving AEs will be followed until resolution, medically stabilized, or 30 days after the study completion/termination visit, whichever comes first. If the severity rating for an ongoing AE changes before the event resolves, the original AE report will be revised (ie, the event will not be reported as separate AE). During the course of any AE, the highest severity rating will be reported.

Deviations from the protocol-specified dosage (including overdosing, underdosing, abuse, and withdrawal, treatment errors (including incorrect route of administration, use of an incorrect product, and deviations from the protocol-defined dosing schedule), failures of expected pharmacological actions, and unexpected therapeutic or clinical

benefits will be followed with regard to occurrence of AEs, lack of efficacy, and/or other observations because these events may be reportable to regulatory authorities.

Any pregnancy that occurs after administration of IP will be reported on a Pregnancy Form and followed-up at 1 year post-delivery, if feasible.

If an investigator becomes aware of an SAE occurring in a subject after study completion, the SAE must be reported on the SAE Form within 24 hours after awareness; no additional reporting on CRFs is necessary.

## **13.2.2.1** Severity

The investigator will assess the severity of each AE using his/her clinical expertise and judgment based on the most appropriate description below:

#### Mild

- The AE is a transient discomfort and does not interfere in a significant manner with the subject's normal functioning level.
- ➤ The AE resolves spontaneously or may require minimal therapeutic intervention.

#### Moderate

- ➤ The AE produces limited impairment of function and may require therapeutic intervention.
- The AE produces no sequela/sequelae.

#### Severe

- ➤ The AE results in a marked impairment of function and may lead to temporary inability to resume usual life pattern.
- ➤ The AE produces sequela/sequelae, which require (prolonged) therapeutic intervention.

These severity definitions will also be used to assess the severity of an AE with a study-related procedure(s), if necessary.

## **13.2.2.2** Causality

Causality is a determination of whether there is a reasonable possibility that the IP is etiologically related to/associated with the AE. Causality assessment includes, eg, assessment of temporal relationships, dechallenge/rechallenge information, association (or lack of association) with underlying disease, presence (or absence) of a more likely cause, and physiological plausibility. For each AE, the investigator will assess the causal

relationship between the IP and the AE using his/her clinical expertise and judgment according to the following most appropriate algorithm for the circumstances of the AE:

- Not related (both circumstances must be met)
  - ➤ Is due to underlying or concurrent illness, complications, concurrent treatments, or effects of concurrent drugs
  - ➤ Is not associated with the IP (ie, does not follow a reasonable temporal relationship to the administration of IP or has a much more likely alternative etiology).
- Unlikely related (either 1 or both circumstances are met)
  - ➤ Has little or no temporal relationship to the IP
  - ➤ A more likely alternative etiology exists
- Possibly related (both circumstances must be met)
  - Follows a reasonable temporal relationship to the administration of IP
  - ➤ An alternative etiology is equally or less likely compared to the potential relationship to the IP
- Probably related (both circumstances must be met)
  - ➤ Follows a strong temporal relationship to the administration of IP, which may include but is not limited to the following:
    - Reappearance of a similar reaction upon re-administration (positive re-challenge)
    - o Positive results in a drug sensitivity test (skin test, etc.)
    - Toxic level of the IP as evidenced by measurement of the IP concentrations in the blood or other bodily fluid
  - ➤ Another etiology is unlikely or significantly less likely

For events assessed as not related or unlikely related, and occurring within 24 hours of IP administration, the investigator shall provide the alternative etiology. These causality definitions will also be used to assess the relationship of an AE with a study-related procedure(s), if necessary.

## 13.3 Urgent Safety Measures

An urgent safety measure is an immediate action taken, which is not defined by the protocol, in order to protect subjects participating in a clinical trial from immediate harm. Urgent safety measures may be taken by the sponsor or clinical investigator, and may include any of the following:

- Immediate change in study design or study procedures
- Temporary or permanent halt of a given clinical trial or trials
- Any other immediate action taken in order to protect clinical trial participants from immediate hazard to their health and safety

The investigator may take appropriate urgent safety measures in order to protect subjects against any immediate hazard to their health or safety. The measures should be taken immediately and may be taken without prior authorization from the sponsor. In the event(s) of an apparent immediate hazard to the subject, the investigator will notify the sponsor immediately by phone and confirm notification to the sponsor in writing as soon as possible, but within 1 calendar day after the change is implemented. The sponsor will also ensure the responsible ethics committee is notified of the urgent measures taken in such cases according to local regulations.

#### 13.4 Untoward Medical Occurrences

Untoward medical occurrences occurring <u>before</u> the first exposure to IP are not considered AEs (according to the definition of AE, see Section 13.2). However, each **serious** untoward medical occurrence experienced <u>before</u> the first IP exposure (ie, from the time of signed informed consent up to but not including the first IP exposure) will be described on the SAE Report. These events will not be considered as SAEs and will not be included in the analysis of SAEs.

For the purposes of this study, each non-serious untoward medical occurrence experienced by a subject undergoing study-related procedures (eg, during blood sampling) <u>before</u> the first IP exposure will be recorded on the AE CRF; these events will not be considered as AEs and will not be included in the analysis of AEs.

## 13.5 Medical Device Safety reporting

The IP kit contains the BAXJECT device. All Serious Injuries (SI) and Unexpected Adverse Device Events (UADE) must be reported. Serious injury is defined as:

• Life-threatening injury or illness results in permanent impairment/ damage to body function/ structure. It requires medical or surgical intervention to preclude permanent impairment/ damage to body function/ structure.

# **13.6 Non-Medical Complaints**

A non-medical complaint (NMC) is any alleged product deficiency that relates to identity, quality, durability, reliability, safety and performance of the product but **did not result in an AE.** NMCs include but are not limited to the following:

- A failure of a product to exhibit its expected pharmacological activity and/or design function, eg, reconstitution difficulty
- Missing components
- Damage to the product or unit carton
- A mislabeled product (eg, potential counterfeiting/tampering)
- A bacteriological, chemical, or physical change or deterioration of the product causing it to malfunction or to present a hazard or fail to meet label claims

Any NMCs of the product will be documented on an NMC form and reported to the sponsor within 1 business day. If requested, defective product(s) will be returned to the sponsor for inspection and analysis according to procedures.

# 13.7 Medical, Medication, and Non-Drug Therapy History

At screening, the subject's medical history will be described for the following body systems including severity (defined in Section 13.2.2.1) or surgery and start and end dates, if known: eyes, ears, nose, and throat; respiratory; cardiovascular; gastrointestinal; musculoskeletal; neurological; endocrine; hematopoietic/lymphatic; dermatological; and genitourinary.

The historical ABR including treated and untreated bleeding episodes in the 12 months prior to study enrollment based on medical records should also be recorded in the eCRF. Only the treated bleeds will be the basis for inclusion in the study.

All medications taken and non-drug therapies received from 4 weeks before enrollment until completion/termination will be recorded on the concomitant medications and non-drug therapies CRFs.

Any prior use of any pegylated medication (name of drug, indication, and dates of use), at any time in the past, will be recorded on the eCRF.

## 13.8 Physical Examinations

At screening and subsequent study visits (as described in the schedule in 21.2), a physical examination will be performed on the following body systems: general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological. At screening, if an abnormal condition is detected, the condition will be described on the medical history CRF. At screening, the Karnofsky performance score will be assessed.

At study visits, if a new abnormal or worsened abnormal pre-existing condition is detected, the condition will be described on the AE CRF. If the abnormal value was not deemed an AE because it was due to an error, due to a preexisting disease (described in Section 13.2.1.4), not clinically significant, a symptom of a new/worsened condition already recorded as an AE, or due to another issue that will be specified, the investigator will record the justification on the source record.

## 13.9 Clinical Laboratory Parameters

All assessments will be performed at a central laboratory, according to the laboratory manual.

At all laboratory assessments subjects must not be actively bleeding. In addition to the laboratory assessments planned in the protocol, appropriate clinical laboratory testing should be performed whenever clinically indicated.

Details on the visits and timing of blood sampling for the laboratory parameters are provided in Supplement 21.2 and Supplement 21.3.

# 13.9.1 Screening Laboratory Parameters

## **13.9.1.1 Blood Type**

For subjects who do not have documentation of their blood type in their medical record, blood ABO blood type will be measured centrally at screening.

## 13.9.1.2 Genetics and HLA-Genotype

FVIII gene mutation analysis and HLA genotype will be analyzed at screening. If results of FVIII gene mutation analysis and HLA genotype are already available at the study site, they will be provided to the sponsor and a reanalysis will not be required in those subjects.

## 13.9.1.3 Pregnancy Test

A pregnancy test should be performed as appropriate (serum pregnancy test in females of child-bearing potential if no urine sample is available). The pregnancy test might be repeated during the study in countries where mandated by national law.

#### 13.9.2 CD4 Count

At screening only, CD4 levels will be determined in all HIV+ subjects using flow cytometry.

## 13.9.3 Viral Serology

Viral serology testing will include HIV-1 and HIV-2 antibody, HBsAb, HBsAg, HBcAb, and HCV Ab. HCV titer will be confirmed by PCR for all subjects reported as HCV positive. All assessments will be performed at screening only. A positive test for HBsAg will be repeated using a new blood sample.

## 13.9.4 Hematology, Clinical Chemistry and Lipid Panel

Hematology tests will be performed on EDTA-anticoagulated whole blood, and clinical chemistry assessments and the lipid panel will be performed on serum.

The hematology panel consists of complete blood count [hemoglobin, hematocrit, erythrocytes (ie, red blood cell count), and leukocytes (ie, white blood cell count)] with differential (ie, basophils, eosinophils, lymphocytes, monocytes, neutrophils), mean corpuscular volume (MCV), mean corpuscular hemoglobin concentration (MCHC), and platelet count.

The clinical chemistry panel consists of sodium, potassium, chloride, bicarbonate, total protein, albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, blood urea nitrogen, creatinine, and glucose.

The lipid panel consists of cholesterol, very low density lipoprotein (VLDL), low density lipoprotein (LDL), high density lipoprotein (HDL) and triglycerides.

## 13.9.5 FVIII Activity, FVIII Antigen, VWF Antigen

Blood samples will be analyzed for FVIII activity (1-stage clotting assay and the chromogenic assay) at a central laboratory. The 1-stage clotting assay will serve as the primary assay; the chromogenic assay will be used to provide supportive data. In addition FVIII antigen will be measured by ELISA. VWF antigen will be determined using ELISA from pre-infusion samples. The detailed time points of FVIII activity, FVIII antigen and VWF antigen assessment are provided in Section 12.1, Section 12.2, and Supplement 21.4.

## 13.9.6 Thrombin Generation Assay

For TGA parameters (lag time, time to peak thrombin generation, peak thrombin generation, and endogenous thrombin potential [ETP]), plasma samples will be tested using the calibrated, automated thrombin generation method (CAT). For details on the individual time points for TGA assessment please see Section 12.1, Supplement 21.2, and Supplement 21.4.

## 13.9.7 Assessment of Laboratory Values

# 13.9.7.1 Assessment of Abnormal Laboratory Values

The investigator's assessment of each laboratory value (ie, hematology, clinical chemistry, and lipids) will be recorded on the CRF. For each abnormal laboratory value, the investigator will determine whether the value is considered clinically significant or not. For clinically significant values, the investigator will indicate if the value constitutes a new AE (see definition in Section 13.2, and record the sign, symptom, or medical diagnosis on the AE CRF), is a symptom or related to a previously recorded AE, is due to a pre-existing disease (described in Section 13.2.1.4), or is due to another issue that will be specified. If the abnormal value was not clinically significant, the investigator will indicate the reason, ie because it is due to a preexisting disease, due to a lab error, or due to another issue that will be specified. Additional tests and other evaluations required to establish the significance or etiology of an abnormal value, or to monitor the course of an AE should be obtained when clinically indicated. Any abnormal value that persists should be followed at the discretion of the investigator.

# 13.9.8 Biobanking

Patients will consent for taking an extra blood sample at each study visit for additional analysis, if necessary. Additional backup samples that remain after study testing is done may be stored and used for additional testing (eg, further evaluation of an abnormal test or an AE). Also, an additional blood draw for exploratory testing will be drawn preinfusion and early in the morning at each study visit, if feasible, otherwise at the same time point at each study visit.

Samples will be stored in a coded form for no more than 2 years after the final study report has been completed and then the samples will subsequently be destroyed.

## 13.10 Vital Signs

Vital signs will include body temperature (°C or °F), respiratory rate (breaths/min), pulse rate (beats/min), and systolic and diastolic blood pressure (mmHg). Height (in or cm) and weight (lb or kg) will also be collected at screening; weight will also be recorded before any IP infusions are administered at the study site, but at least at each study visit. Blood pressure will be measured when subjects are in the supine position.

Vital signs will be assessed within 15 minutes prior to start of infusion and 30±5 minutes following infusion at baseline and at each study visit. Vital signs should always be assessed before any blood sampling is done at a particular time point.

Vital sign values are to be recorded on the CRF. For each abnormal vital sign value, the investigator will determine whether or not to report an AE (see definition in Section 13.2 and record the medical diagnosis (preferably), symptom, or sign on the AE CRF). Additional tests and other evaluations required to establish the significance or etiology of an abnormal value, or to monitor the course of an AE should be obtained when clinically indicated. Any abnormal value that persists should be followed at the discretion of the investigator.

#### 14. STATISTICS

# 14.1 Sample Size and Power Calculations

## 14.1.1 Sample Size Calculation

For the sample size assessment the following assumptions were used. Approximately 40% of patients in BAX 855 regimen targeting 1-3% trough level are expected to be bleed-free as shown in the ADVATE Prophylaxis study and the BAX 855 pivotal study 261201. For the BAX 855 regimen targeting approximately 10% (8-12%) trough level, an increase to 70% bleed-free patients is expected based on modeling the bleeding rates per factor VIII level in the BAX 855 pivotal study 261201.

Under these assumptions 48 subjects per study arm are needed to reject the null hypothesis of no difference between the study arms against a two-sided alternative at the 5% level of statistical significance with 80% power. Assuming a drop-out rate of close to 10%, and 10-15% of subjects being non-compliant, approximately 116 subjects are planned to be randomized between the two BAX 855 regimens with an allocation ratio of 1:1.

## 14.2 Datasets and Analysis Cohorts

#### 14.2.1 Full Analysis Set

The Full Analysis Set (FAS) will comprise all subjects who were randomized and who were treated with BAX 855 prophylactically for any period of time.

#### 14.2.2 Per Protocol Analysis Set

The Per Protocol Analysis Set will comprise all subjects who were randomized and completed the second 6 months of prophylactic treatment.

#### 14.2.3 Safety Analysis Set

The Safety Analysis Set (SAS) will comprise all subjects treated with at least 1 BAX 855 dose. All safety analyses for BAX 855 will be performed on the SAS.

## 14.3 Handling of Missing, Unused, and Spurious Data

Missing data will not be imputed in general, with the exceptions as detailed below.

## 14.3.1 Handling of incomplete observation periods for ABR

The primary endpoint requires complete data for the second 6 months of prophylaxis (Day 184 to Day 366). The multiple imputations technique will be used for the analysis of the primary endpoint and estimation of ABRs. As this is a statistical analysis technique, it will be described in the statistical analysis section.

## 14.3.2 Handling of other variables

If body weight is missing for a subject then the last value of available body weight measurement will be carried forward in order to compute weight-adjusted BAX 855 consumption. If the date of onset for an AE is missing completely then it will be imputed with the date of the first study drug application.

For PK data, if any concentration data are considered spurious (e.g. lack of biological plausibility), the reason for exclusion and the analysis from which the data point was excluded will be documented.

Regarding missing data in AE records:

- Handling of unknown causality assessment:
  - ➤ If a subject experiences an AE with a missing causality assessment, the relationship of the AE will be counted as "related".
- Handling of unknown severity grades:
  - ➤ If a subject experiences more than one AE categorized under the same preferred term, one of them is categorized as "severe" and one of them is categorized as "unknown", the severity of this AE will be counted as "severe".
- If a subject experiences more than one AE categorized under the same preferred term, one of them is categorized as "mild" or "moderate" and one of them is categorized as "unknown", the severity of this AE will be counted as "unknown".

#### 14.4 Methods of Analysis

## 14.4.1 Primary Outcome Measure

The proportion of subjects with ABR = 0 in the two prophylaxis treatment regimens in the second 6 months period will be compared using a chi-square test with continuity correction at a two-sided 5% level of significance.

The null hypotheses of no difference between the prophylactic regimens will be tested against a two-sided alternative.

The observation period for the primary endpoint will be the second 6 months of prophylaxis (Day 184 to Day 366). If the subject undergoes a surgical procedure the observation period is interrupted starting from the presurgical loading dose until the subject resumes his previous prophylactic treatment regimen, or until rehabilitation or any other surgery specific postoperative measures have been completed, whichever occurs last.

The multiple imputations (MI) technique will be used to handle observation periods shorter than 6 months, i.e. 183 days, as follows.

For subjects who terminated before Day 366, bleeds will be imputed for the unobserved period from a Poisson random variate. The subject specific Poisson parameter will be determined from estimating a negative binomial model for the bleed rate in the unobserved period with stratum, age, race as well as the number of bleeds in the observed period of the subject as covariates in all subjects of the same Study Arm. For subjects with more than 150 days in the observation period, the number of bleeds occurring at a later time in other subjects might be very low or even zero. To avoid estimating from an unstable model, the negative binomial model will be for the number of bleed up to Day 150 with covariates of stratum, age, race and number of bleeds observed up to Day 150. At least 1000 imputation datasets will be generated. The chi-squared test statistics with continuity correction and its standard error will be used to compare the two study arms in each imputation dataset and the multiple imputations techniques will be used to derive an overall estimate with two-sided 95% confidence interval.

The dataset to be analyzed is all subjects with any observation time between Day 184 and 366 and all subjects who developed an inhibitor (at any time); the latter being considered to have had a bleed.

The use of age and race in the imputation model will allow for subgroup analyses of the primary endpoint and ABRs.

Sensitivity analyses

Sensitivity analyses will be performed similar to the primary analysis except that the negative binomial distributions used for imputations will have an artificially increased Poisson parameter by 10%, 20% and 30%.

## 14.4.2 Secondary Outcome Measures

• Spontaneous and traumatic ABR, and spontaneous AJBR

For total ABR, spontaneous ABR, traumatic ABR and spontaneous JABR, separate negative binomial models will be used for the second 6 months treatment period.

The negative binomial model for the bleed rate with covariates of Study Arm, stratum, age, and race. The multiple imputations technique will be used for incomplete observation periods as described for the primary endpoints analysis. Subgroups for age and race will be analyzed as well.

For all other outcome measures, descriptive statistics will be presented for the two dosing regimens. Point estimates (means and medians) and their 95% CIs will be computed to include:

- Total weight-adjusted consumption of BAX 855 for each prophylactic regimen
- Overall hemostatic efficacy rating at  $24 \pm 2$  h after initiation of treatment and at resolution of bleed
- Number of BAX 855 infusions needed for the treatment of bleeding episodes
- HJHS
- Physical domain and component scores of the SF-36
- Physical Activity Levels

In case of surgeries, descriptive statistics will be performed for the following secondary outcome measures:

• Intra-, post- and perioperative hemostatic efficacy in case of surgery

Intra- and postoperative blood loss in case of surgery

PK parameters before randomization will be summarized descriptively over all subjects to include:

 $AUC_{0-\infty}$  (Area under the plasma concentration versus time curve from time 0 to infinity), IR (incremental recovery) at 15-30 minutes post-infusion,  $T_{1/2}$  (plasma half-life), MRT (mean residence time), CL (clearance), maximum plasma concentration (Cmax) and time to maximum concentration in plasma (Tmax),  $V_{ss}$  (Volume of distribution at steady state)

PK parameters after 9 months will be summarized descriptively by prophylactic treatment regimen:

 $AUC_{0-\infty}$  (Area under the plasma concentration versus time curve from time 0 to infinity), IR (incremental recovery) at 15-30 minutes post-infusion,  $T_{1/2}$  (plasma half-life), CL (clearance), maximum plasma concentration (Cmax) and time to maximum concentration in plasma (Tmax),

Incremental recovery (IR) over time will be displayed as boxplots for the two prophylactic regimens.

Correlation of VWF:Ag and PK parameters will be assessed by boxplots and Spearman rank correlation coefficient.

Descriptive statistics will be used for the secondary safety outcome measures (see Section 8.4.2.2):

- Occurrence of AEs and SAEs
- Changes in vital signs and clinical laboratory parameters (hematology, clinical chemistry, and lipids)
- Inhibitory antibodies to FVIII, and binding antibodies to FVIII, BAX 855, PEG, and CHO protein

The methods of analysis for the secondary PROs measures (see Section 8.4.2.3) are described for the following PROs:

- Physical domain and component scores of the SF-36
- Physical activity levels

Change scores from baseline to completion/follow-up will be assessed for each treatment arm and tested using the minimally important difference threshold and the Wilcoxon sign rank test. Differences in the change scores between treatment groups will be tested using the minimally importance difference threshold and the Mann-Whitney U Test.

# **14.4.3 Exploratory Outcome Measures**

Boxplots and Spearman rank correlation coefficient will be used to assess the correlation between the average of various coagulation parameters (thrombin generation assay (TGA) parameters: lag time, time to peak thrombin generation, peak thrombin generation, and endogenous thrombin potential [ETP] and FVIII trough levels) and ABR in the same time periods (first 6 months, second 6 months, overall).

Changes from baseline to completion/follow-up for patients for the two dosing arms will be tested using the minimally importance difference threshold and the Wilcoxon sign rank test for the following PROs:

- Bleed and pain severity as measured by the Haemo-SYM questionnaire
- HRQoL as assessed using the EQ-5D and mental domain and component scores of the SF-36 questionnaire
- Health Resource Utilization

Differences in the change scores between treatment groups will be tested using the minimally importance difference threshold and the Mann-Whitney U Test for the following PROs:
- Bleed and pain severity as measured by the Haemo-SYM questionnaire
- HRQoL as assessed using the EQ-5D and mental domain and components scores of the SF-36 questionnaire
- Health Resource Utilization

# 15. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

The investigator/study site will cooperate and provide direct access to study documents and data, including source documentation for monitoring by the study monitor, audits by the sponsor or sponsor's representatives, review by the EC, and inspections by applicable regulatory authorities, as described in the Clinical Study Agreement. If contacted by an applicable regulatory authority, the investigator will notify the sponsor of contact, cooperate with the authority, provide the sponsor with copies of all documents received from the authority, and allow the sponsor to comment on any responses, as described in the Clinical Study Agreement.

## 16. QUALITY CONTROL AND QUALITY ASSURANCE

# 16.1 Investigator's Responsibility

The investigator will comply with the protocol (which has been approved/given favorable opinion by the EC), ICH GCP, and applicable regulatory requirements as described in the Clinical Study Agreement. The investigator is ultimately responsible for the conduct of all aspects of the study at the study site and verifies by signature the integrity of all data transmitted to the sponsor. The term "investigator" as used in this protocol as well as in other study documents, refers to the investigator or authorized study personnel that the investigator has designated to perform certain duties. Sub-investigators or other authorized study personnel are eligible to sign for the investigator, except where the investigator's signature is specifically required.

# **16.1.1 Final Clinical Study Report**

The investigator, or coordinating investigator(s) for multicenter studies, will sign the clinical study report. The coordinating investigator will be selected before study start.

# 16.2 Training

The study monitor will ensure that the investigator and study site personnel understand all requirements of the protocol, the investigational status of the IP, and his/her regulatory responsibilities as an investigator. Training may be provided at an investigator's meeting, at the study site, and/or by instruction manuals. In addition, the study monitor will be available for consultation with the investigator and will serve as the liaison between the study site and the sponsor.

#### 16.3 Monitoring

The study monitor is responsible for ensuring and verifying that each study site conducts the study according to the protocol, standard operating procedures, other written instructions/agreements, ICH GCP, and applicable regulatory guidelines/requirements. The investigator will permit the study monitor to visit the study site at appropriate intervals, as described in the Clinical Study Agreement. Monitoring processes specific to the study will be described in the clinical monitoring plan.

#### 16.4 Auditing

The sponsor and/or sponsor's representatives may conduct audits to evaluate study conduct and compliance with the protocol, standard operating procedures, other written instructions/agreements, ICH GCP, and applicable regulatory guidelines/requirements. The investigator will permit auditors to visit the study site, as described in the Clinical Study Agreement. Auditing processes specific to the study will be described in the auditing plan.

# **16.5 Non-Compliance with the Protocol**

The investigator may deviate from the protocol only to eliminate an apparent immediate hazard to the subject. In the event(s) of an apparent immediate hazard to the subject, the investigator will notify the sponsor immediately by phone and confirm notification to the sponsor in writing as soon as possible, but within 1 calendar day after the change is implemented. The sponsor will also ensure the responsible ethics committee is notified of the urgent measures taken in such cases according to local regulations.

If monitoring and/or auditing identify serious and/or persistent non-compliance with the protocol, the sponsor may terminate the investigator's participation. The sponsor will notify the EC and applicable regulatory authorities of any investigator termination.

# 16.6 Laboratory and Reader Standardization

Not applicable; a central laboratory will be used for all clinical assessments.

#### **17. ETHICS**

# 17.1 Subject Privacy

The investigator will comply with applicable subject privacy regulations/guidance as described in the Clinical Study Agreement.

# 17.2 Ethics Committee and Regulatory Authorities

Before enrollment of patients into this study, the protocol, informed consent form, any promotional material/advertisements, and any other written information to be provided will be reviewed and approved/given favorable opinion by the EC and applicable regulatory authorities. The IB will be provided for review. The EC's composition or a statement that the EC's composition meets applicable regulatory criteria will be documented. The study will commence only upon the sponsor's receipt of approval/favorable opinion from the EC and, if required, upon the sponsor's notification of applicable regulatory authority(ies) approval, as described in the Clinical Study Agreement.

If the protocol or any other information given to the subject is amended, the revised documents will be reviewed and approved/given favorable opinion by the EC and applicable regulatory authorities, where applicable. The protocol amendment will only be implemented upon the sponsor's receipt of approval and, if required, upon the sponsor's notification of applicable regulatory authority(ies) approval.

#### 17.3 Informed Consent

Investigators will choose patients for enrollment considering the study eligibility criteria. The investigator will exercise no selectivity so that no bias is introduced from this source.

All patients and/or their legally authorized representative must sign an informed consent form before entering into the study according to applicable regulatory requirements and ICH GCP. An assent form may be provided and should be signed by patients less than 18 years of age. Before use, the informed consent/assent form will be reviewed by the sponsor and approved by the EC and regulatory authority(ies), where applicable, (see Section 17.2). The informed consent/assent form will include a comprehensive explanation of the proposed treatment without any exculpatory statements, in accordance with the elements required by ICH GCP and applicable regulatory requirements. Patients and/or their legally authorized representative(s) will be allowed sufficient time to consider participation in the study. By signing the informed consent/assent form, patients and/or their legally authorized representative(s) agree that they will complete all evaluations required by the study, unless they withdraw voluntarily or are terminated from the study for any reason.

The sponsor will provide to the investigator in written form any new information that significantly bears on the subjects' risks associated with IP exposure. The informed consent/assent will be updated, if necessary. This new information and/or revised informed consent/assent form that have been approved by the applicable EC and regulatory authorities, where applicable, will be provided by the investigator to the subjects and/or the subjects' legally authorized representative who consented to participate in the study (see Section 17.3).

# 17.4 Data Monitoring Committee

A Data Monitoring Committee (DMC) will not be used for this study as the expected related AEs in this study are anticipated to be similar to that of the licensed product ADVATE (of which the core protein is identical to that of BAX 855; see Section 6.5 for more details on anticipated risks and benefits of BAX 855). Additionally, the safety is not expected to differ from the safety observed in the BAX 855 pivotal and the ongoing BAX855 continuation study (Studies 261201 and 261302, respectively).

#### 18. DATA HANDLING AND RECORD KEEPING

# **18.1 Confidentiality Policy**

The investigator will comply with the confidentiality policy as described in the Clinical Study Agreement.

# 18.2 Study Documentation and Case Report Forms

The investigator will maintain complete and accurate paper format study documentation in a separate file. Study documentation may include information defined as "source data" (see Section 8.8), records detailing the progress of the study for each subject, signed informed consent forms, correspondence with the EC and the study monitor/sponsor, enrollment and screening information, CRFs, SAE reports (SAERs), laboratory reports (if applicable), and data clarifications requested by the sponsor.

The investigator will comply with the procedures for data recording and reporting. Any corrections to paper study documentation must be performed as follows: 1) the first entry will be crossed out entirely, remaining legible; and 2) each correction must be dated and initialed by the person correcting the entry; the use of correction fluid and erasing are prohibited.

The investigator is responsible for the procurement of data and for the quality of data recorded on the CRFs. CRFs will be provided in electronic form.

If electronic format CRFs are provided by the sponsor, only authorized study site personnel will record or change data on the CRFs. If data is not entered on the CRFs during the study visit, the data will be recorded on paper, and this documentation will be considered source documentation. Changes to a CRF will require documentation of the reason for each change. An identical (electronic/paper) version of the complete set of CRFs for each subject will remain in the investigator file at the study site in accordance with the data retention policy (see Section 18.3).

The handling of data by the sponsor, including data quality assurance, will comply with regulatory guidelines (eg, ICH GCP) and the standard operating procedures of the sponsor. Data management and control processes specific to the study will be described in the data management plan.

# 18.3 Document and Data Retention

The investigator will retain study documentation and data (paper and electronic forms) in accordance with applicable regulatory requirements and the document and data retention policy, as described in the Clinical Study Agreement.

# 19. FINANCING AND INSURANCE

The investigator will comply with investigator financing, investigator/sponsor insurance, and subject compensation policies, if applicable, as described in the Clinical Study Agreement.

# **20. PUBLICATION POLICY**

The investigator will comply with the publication policy as described in the Clinical Study Agreement.

# **21. SUPPLEMENTS**

# **21.1 Study Flow Charts**

Figure 1
Study Design for Baxalta Clinical Study 261303



PHA = Patient with severe Hemophilia A

PK = Assessment of individual PK parameters

R = Randomization



<sup>\*</sup> Washout: Low trough arm: 96 h (after the longer treatment interval of 4 days), 72 h (after the short treatment interval of 3 days) or 84 h (3.5 day intervals); High trough arm: at least 48 h or when the subject reaches his/her baseline value.

# 21.2 Detailed Flow Diagram of Study Procedures

Before **any** study procedures are performed, informed consent must be obtained from each patient.

# **Screening Visit**

The screening procedures differ according to whether the subject is **transitioning from a previous BAX 855 study** (see Section A) or is newly recruited (see Section B). If the sponsor decides a transitioning subject requires a PK Assessment, then from the screening visit onwards procedures are identical to those for newly recruited subjects. If no PK Assessment is required, the next visit for transitioning subjects is the Baseline Visit once randomization is performed.

Evaluations must be completed within 56 days of the screening visit.

No wash-out is required but whenever possible the screening visit should be scheduled shortly before the next scheduled prophylactic infusion when baseline FVIII trough levels are reached in case the subject receives prophylactic treatment.

#### A: Subjects transitioning from other BAX 855 studies

The screening visit coincides with the end of study visit of the previous BAX 855 study; the subject must not be actively bleeding. If applicable, BAX 855 will be administered for IR determination based on the protocol of the previous study.

Informed consent must be obtained at enrollment at the latest (prior to any study-specific procedure); to give the patient sufficient time to review the ICF, this document should preferably be provided prior to the end of study visit of the previous study.

The relevant data obtained at the end of study visit of the previous BAX 855 study will be transcribed to the screening visit eCRF of this PK-guided dosing study, and where possible, duplication of blood draws or evaluations will be avoided.

The following procedures will be performed:

#### **Clinical Assessments:**

- Assessment of inclusion/exclusion criteria
- PROs (or can be done at Baseline visit) should be determined prior to any other study specific procedures:
  - Haemo-SYM questionnaire
  - o EO-5D
  - o SF-36
  - Physical activity questionnaire
  - Health Resource Use

#### **Laboratory Assessments:**

Blood will be drawn for the following additional assessments:

- Screening tests:
  - CD4 count in subjects who are HIV positive
  - O Viral serology (if any positive, test to be confirmed with a second sample):
    - HIV: HIV-1 and HIV-2 Ab
    - HBV: HBsAg, HBsAb, HBcAb
    - HCV: HCVAb (PCR to be performed if positive)
- · Pregnancy test, if applicable

The following data will be obtained/transcribed from the end of study visit of the previous BAX 855 study:

- · Medical history
- Medication history
- Concomitant medications
- · Non-drug therapies
- Physical examination (including assessment of target joints)
- Vital signs (body temperature (°C), respiratory rate (breaths/min), pulse rate (beats/min), and supine systolic and diastolic blood pressure (mmHg)).
- Laboratory Data:
  - o FVIII/VWF/TGA assays:
    - FVIII activity (activated partial thromboplastin-based 1-stage clotting assay and chromogenic assay)
    - FVIII antigen
    - VWF antigen
    - TGA, if not available from previous study, an additional blood sample has to be drawn for TGA testing
  - o Immunogenicity tests:
    - Inhibitory antibodies to FVIII (Nijmegen assay)
    - Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
    - Anti-CHO antibodies
  - o Hematology, clinical chemistry, and lipids
  - o Gene mutation and HLA genotype if not available
  - o Blood type (A, B, AB or O) if historical data not available

#### Subject diary:

• Hand out subject diary and provide training to subject

## Other procedures:

- Dispense IP:
  - A sufficient quantity of IP of study 261303 will be dispensed to cover the period until the PK Assessment / Baseline visit (as applicable)

#### **B:** Newly recruited subjects

- Ensure informed consent has been obtained
- Medical history
- Hemophilia history, including:
  - Confirmation of diagnosis and severity
  - o Family history of hemophilia
  - o Documentation of mutation, if known
  - The presence of any target joints will be documented. A target joint is defined as any single joint (ankles, knees, hips, or elbows) with  $\geq 4$  spontaneous bleeding episodes in any consecutive 6 month period.
  - o Documentation of all FVIII replacement therapies used within the last year, including:
    - Date of last FVIII infusion prior to screening visit, type of FVIII product, dose infused and reason for administration
    - FVIII regimen (prophylaxis or on-demand)
    - Product name (or IP name and manufacturer, if applicable)
    - Dose (for prophylaxis, if applicable, and for treatment of bleeding episodes)
    - Frequency of administration (for prophylaxis)

- Estimate of average number of infusions for each bleeding episode and usual response
- Assessment of subject's ABR based on documented and treated bleeding episodes within 12 months before enrolment, based on subject's medical records.
- Concomitant medications for the last 30 days, and any prior history of use of any pegylated medication (eg, PEG-interferon) at any time in the past, including treatment indication, date of last administration, and duration of treatment(s), if known
- Non-drug therapies for the last 30 days
- Physical examination, including height and weight
- Karnofsky performance score
- Vital signs (body temperature (°C), respiratory rate (breaths/min), pulse rate (beats/min), and supine systolic and diastolic blood pressure (mmHg)).
- PROs (or can be done at Baseline visit) should be determined before any other study specific procedures are performed:
  - Haemo-SYM questionnaire
  - o EQ-5D
  - o SF-36
  - Physical activity questionnaire
  - o Health Resource Use

#### **Laboratory Assessments:**

Blood will be drawn for the following assessments:

- Screening tests:
  - o CD4 count in subjects who are HIV positive
  - O Viral serology (if any positive, test to be confirmed with a second sample):
    - HIV: HIV-1 and HIV-2 Ab
    - HBV: HBsAg, HBsAb, HBcAb
    - HCV: HCVAb (PCR to be performed if positive)
  - Genetics (FVIII gene mutation analysis) and HLA-genotype if historical data not available
  - o Blood type (A, B, AB or O) if historical data not available
- FVIII/VWF/TGA assays:
  - FVIII activity (activated partial thromboplastin-based 1-stage clotting assay and chromogenic assay)
  - o FVIII antigen
  - o VWF antigen
  - o TGA
- Immunogenicity tests:
  - o Inhibitory antibodies to FVIII (Nijmegen assay)
  - o Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
  - Anti-CHO antibodies
- Hematology, clinical chemistry, and lipids
- Pregnancy test, if applicable

#### Subject diary:

Hand out subject diary and provide training to subject

#### **PK** Assessment

Subjects transitioning from another BAX 855 study who have already had a PK assessment may have to repeat the PK assessment based on the sponsor's evaluation. The PK assessment has to be performed after a wash-out period of at least 72-96 h depending on the FVIII concentrate used and the patient should not be actively bleeding.

Blood sampling after infusion of BAX 855 for PK assessments will be performed over a 4-day period.

• Review and discuss subject diary

At the **pre-infusion** time point, the following assessments will be carried out:

- Laboratory Assessments (within 30 minutes of start of infusion):
  - FVIII assays
  - o VWF antigen
  - o TGA
- Vital signs (within 15 minutes of start of infusion)

#### Infusion:

• Infusion of  $60 \pm 5$  IU/kg BAX 855

#### Post-infusion:

- Laboratory Assessments:
  - FVIII assays and TGA at the post-infusion time points, 15-30 min, 3±0.5 h, 8±0.5 h, 24±2 h, 48±2 h, 72±4 h and 96±4 h

At  $30 \pm 5$  min post-infusion:

• Vital signs (body temperature, respiratory rate, pulse rate, and supine systolic and diastolic blood pressure)

**Throughout the visit**, the following assessments will be carried out:

- Physical examination
- Adverse events
- Concomitant medications and non-drug therapies

#### Randomization

Once the FVIII activity results are available and the PK parameters calculated, subjects will be randomized to one of the treatment arm.

#### **Baseline Visit**

The washout periods are at least 72 - 96 h and the subject must not be actively bleeding. Evaluations must be completed within 56 days of the PK Assessment. Whenever possible the PRO questionnaires should be completed before all other study specific procedures are started.

At the **pre-infusion** time point, the following assessments will be carried out:

- PROs (if not done at Screening visit):
  - Haemo-SYM questionnaire
  - o EQ-5D
  - o SF-36
  - Physical Activity questionnaire
  - o Health Resource Use
- Review and discuss subject diary
- Physical examination, including body weight, and assessment of target joints
- Vital signs (within 15 minutes of start of infusion)
- Laboratory Assessments (within 30 minutes before start of infusion):
  - o Hematology, clinical chemistry, and lipids
  - o FVIII, VWF Ag and TGA assays
  - o Immunogenicity tests (:
    - Inhibitory antibodies to FVIII (Nijmegen assay)
    - Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
    - Anti-CHO antibodies

#### Infusion:

• Infusion of PK-guided dose of BAX 855

#### **Post-infusion**:

At 15-30 min post-infusion:

- Laboratory Assessments
  - o FVIII and TGA assays

At 30±5 min post infusion:

• Vital signs (body temperature, respiratory rate, pulse rate, and supine systolic and diastolic blood pressure)

#### Other procedures:

- Dispense IP
- HJHS joint score

**Throughout the visit**, the following assessments will be carried out:

- Adverse events
- Concomitant medications and non-drug therapies

# **Visits at Study Site:**

3 months  $\pm$  2 weeks 6 months  $\pm$  2 weeks

For the procedures at 4 weeks  $\pm 5$  days, 8 weeks  $\pm 1$  week and 4.5 months  $\pm 2$  weeks, see next section.

The procedures listed here will also be carried out at 7.5 months  $\pm$  2 weeks and 10.5 months  $\pm$  2 weeks if subject has bleeding and attends site rather than having a phone visit.

The washout periods are as follows: Low trough arm: 96 h (after the longer treatment interval of 4 days), 72 h (after the short treatment interval of 3 days) or 84 h (3.5 day intervals); High trough arm: at least 48 h or when the subject reaches his/her baseline value depending on the frequency of BAX 855 infusions.

The subject must not be actively bleeding.

Before any other study-specific procedures are carried out:

- PROs at 6 month visit
  - o Haemo-SYM questionnaire
  - o EQ-5D
  - o SF-36
  - o Physical Activity
  - Health Resource Use
- EQ-5D, Patient Activity Level, and Health Resource Use at each visit
- Physical examination, including body weight, and assessment of target joints
- Review and discuss subject diary

Re-evaluation of PK regimen based on pre-dose FVIII trough level from previous visit, change in body weight. Note: before any dose adjustments are performed an additional visit should be scheduled within 14 days after receipt of the FVIII activity result to reassess trough levels.

# At the **pre-infusion** time point:

- Vital signs (within 15 minutes of start of infusion)
- Laboratory Assessments (within 30 minutes before start of infusion):
  - Hematology, clinical chemistry, and lipids (clinical chemistry and lipids are not applicable at study visits 7.5 month  $\pm 2$  weeks and 10.5 month  $\pm 2$  weeks)
  - o FVIII, VWF Ag and TGA assays
  - o Immunogenicity tests:
    - Inhibitory antibodies to FVIII (Nijmegen assay)
    - Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
    - Anti-CHO antibodies

#### Infusion:

• Infusion of 60±5 IU/kg of BAX 855

#### **Post-infusion**:

At 15-30 min post-infusion:

• FVIII and TGA assays

At 30±5 min post-infusion:

• Vital signs (body temperature, respiratory rate, pulse rate, and supine systolic and diastolic blood pressure)

#### Dispense IP

**Throughout the visit**, the following assessments will be carried out:

- Adverse events
- Concomitant medications and non-drug therapies

# **Visits at Study Site:**

4 weeks ± 5 days 8 weeks ± 1 week 4.5 months ± 2 weeks Dose Readjustment Visit Visits following dose adjustment

The washout periods are as follows: Low trough arm: 96 h (after the longer treatment interval of 4 days), 72 h (after the short treatment interval of 3 days) or 84 h (3.5 day intervals); High trough arm: at least 48 h or when the subject reaches his/her baseline value, depending on the frequency of BAX 855 infusions.

The subject must not be actively bleeding.

These procedures will also be followed if a subject attends an additional visit to check trough FVIII levels prior to any dose readjustment.

Before any other study-specific procedures are carried out:

- EQ-5D, Patient Activity Level and Health Resource Use
- Review and discuss subject diary
- Re-evaluation of FVIII regimen based on pre-dose FVIII trough level from previous visit, if applicable, change in body weight. Note: before any dose adjustments are performed an additional visit should be scheduled in 14 days to reassess trough levels

At the **pre-infusion** time point, the following assessments will be carried out:

- Vital signs (within 15 minutes of start of infusion)
- Laboratory Assessments:
  - o FVIII, VWF Ag and TGA assays (within 30 minutes of start of infusion)
- Immunogenicity tests (within 30 minutes of start of infusion):
  - o Inhibitory antibodies to FVIII (Nijmegen assay)
  - o Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
  - Anti-CHO antibodies

#### Infusion:

• Infusion of PK-guided dose of BAX 855

## FVIII trough level measurement following dose adjustment

Those subjects who had dose adjustment will undergo a repeat FVIII trough level measurement approximately 2 weeks following their dose adjustment. The measurement should be performed immediately prior to their next scheduled prophylactic infusion:

Only the following assessment will be performed:

- Laboratory Assessments:
  - o FVIII, VWF Ag and TGA assays (within 30 minutes of start of infusion)

**Throughout the visit**, the following assessments will be carried out:

- · Adverse events
- Concomitant medications and non-drug therapies

#### IP dispense

#### **Phone Visits:**

7.5 months  $\pm$  2 weeks 10.5 months  $\pm$  2 weeks

If subject experienced bleeding episodes between the last visit and visit 7.5 months $\pm$  2 weeks and 10.5 months  $\pm$  2 weeks, respectively visits they must attend site rather than having a phone visit

The subject will be contacted by phone and will be asked about the following:

- Review and discuss subject diary
- Bleeding episodes and their treatment
- Adverse events
- Concomitant medications and non-drug therapies

In case of bleeding episodes the following laboratory assessment may be performed (see also procedures for study visit months  $3 \pm 2$  weeks and  $6 \pm 2$  weeks ):

- FVIII, VWF, TGA assay
- Hematology
- IR
- Immunogenicity

Before any study specific procedures:

• EQ-5D, Patient Activity Level, and Health Resource Use

# **Visits at Study Site:**

#### 9 months $\pm$ 2 weeks

The washout periods are as follows:

- Low trough arm: at least 96 h (after the longer treatment interval of 4 days), 72 h (after the short treatment interval of 3 days) or 84 h (3.5 day intervals); prior to the subsequent prophylactic infusion
- High trough arm: at least 48 h immediately prior to next prophylactic infusion or when the subject reaches his/her baseline value depending on the frequency of BAX 855 infusions.

The subject must not be actively bleeding.

Before any other study-specific procedures are carried out:

- EQ-5D, Patient Activity Level, and Health Resource Use
- Review and discuss subject diary

Physical examination, including body weight, and Assessment of target joints

At the **pre-infusion** time point, the following assessments will be carried out:

- Vital signs (within 15 minutes of start of infusion)
- Laboratory Assessments (within 30 minutes of start of infusion):
  - o FVIII, VWF Ag and TGA assays
- Immunogenicity tests (within 30 minutes of start of infusion):
  - o Inhibitory antibodies to FVIII (Nijmegen assay)
  - o Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
  - o Anti-CHO antibodies

#### Infusion:

• Infusion of 60±5 IU/kg BAX 855

#### **Post-infusion**:

- Laboratory Assessments:
  - $\circ$  FVIII assays and TGA at the post-infusion time points, 15-30 min, 3±0.5 h, 8±0.5 h, 24±2 h, 48±2 h, 72±4 h and 96±4 h
  - At  $30 \pm 5$  min post-infusion:
- Vital signs (body temperature, respiratory rate, pulse rate, and supine systolic and diastolic blood pressure)

# **Dispense IP**

Throughout the visit, the following assessments will be carried out:

- Adverse events
- Concomitant medications and non-drug therapies

# **Completion/Termination Visit:**

#### at 12 months $\pm$ 2 weeks

The washout periods are as follows: Low trough arm: at least 96 h (after the longer treatment interval of 4 days), 72 h (after the short treatment interval of 3 days) or 84 h (3.5 day intervals); High trough arm: at least 48 h or when the subject reaches his/her baseline value depending on the frequency of infusions.

The subject must not be actively bleeding.

**Before** any other study-specific procedures are carried out:

- PROs:
  - o Haemo-SYM questionnaire
  - o SF-36
  - o EO-5D
  - o Physical Activity
  - Health Resource Use
- Return of subject diary and review and discuss entries with subject
- Physical examination, including body weight Assessment of target joints HJHS joint score

At the **pre-infusion** time point, the following assessments will be carried out:

- Vital signs (within 15 minutes of start of infusion)
- Laboratory Assessments:
  - o FVIII, VWF Ag and TGA assays (within 30 minutes of start of infusion)
- Immunogenicity tests (within 30 minutes of start of infusion):
  - o Inhibitory antibodies to FVIII (Nijmegen assay)
  - o Binding antibodies (IgG and IgM) to FVIII, BAX 855, and PEG
  - o Anti-CHO antibodies

#### Infusion:

• Infusion of  $60 \pm 5 \text{ IU/kg BAX } 855$ 

#### **Post-infusion**:

- Laboratory Assessments:
  - o FVIII assays and TGA (15-30 minutes after start of infusion)

At  $30 \pm 5$  min post-infusion:

• Vital signs (body temperature, respiratory rate, pulse rate, and supine systolic and diastolic blood pressure)

#### Throughout the visit, the following assessments will be carried out:

- Adverse events
- Concomitant medications and non-drug therapies

# 21.3 Schedule of Study Procedures and Assessments

| | sit | PK Assessment <sup>a</sup> Pre infusion, | it | | | | Study | Visits | | | | Completion/ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures/<br>Assessments | Screening Visit | 15-30 min, 3±0.5 h,<br>8±0.5 h, 24±0.5 h<br>48±2 h, 72±4 h<br>& 96±4 h<br>Post- Infusion | Baseline Visit | Visit<br>4Wk<br>±5d | Visit<br>8Wk<br>±1Wk | Visit<br>3 Mo<br>±2Wk | Visit<br>4.5 Mo<br>±2Wk | Visit<br>6 Mo<br>±2Wk | Phone<br>Visit 7.5<br>Mo<br>±2Wk <sup>b</sup> | Visit<br>9 Mo<br>±2Wk<br>+ PK | Phone<br>Visit<br>10.5 Mo<br>±2wk <sup>b</sup> | Completion/<br>Termination<br>Visit <sup>c</sup><br>12 Mo ±2Wk |
| Washout | N/A | 72-96 h | | | | | | | | | | ment interval of<br>her baseline value |
| Informed consent <sup>d</sup> | X | | | | | | | | | | | |
| Eligibility criteria | X | | | | | | | | | | | |
| Medical and medication history <sup>e</sup> | X* | | | | | | | | | | | |
| Concomitant medications <sup>f</sup> | X* | X | X | X | X | X | X | X | X | X | X | X |
| Non-drug therapies <sup>f</sup> | X* | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>g</sup> | X* | X | X | | | X | | X | $(X)^b$ | X | $(X)^b$ | X |
| Vital signs <sup>h</sup> | X* | X | X | X | X | X | X | X | $(X)^b$ | X | $(X)^b$ | X |
| Adverse events <sup>f</sup> | * | X | X | X | X | X | X | X | X | X | X | X |
| Bleeding episodes and their treatment <sup>f,i</sup> | * | | | X | X | X | X | X | X | X | X | X |
| Assessment of target joints <sup>j</sup> | X | | X | | | X | | X | (X) | X | (X) | X |
| Joint score (HJHS) | | | X | | | | | | | | | X |
| Subject diary <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Laboratory assessments <sup>1</sup> | X* | X | X | X | X | X | X | X | $(X)^{b}$ | X | $(X)^b$ | X |
| IP treatment <sup>m</sup> | | X | X | X | X | X | X | X | $(X)^b$ | X | $(X)^b$ | X |
| IP dispense <sup>n</sup> | X <sup>n</sup> | (X) | X | X | | X | | X | | X | | |
| Re-evaluation of PK regimen/dose adjustments <sup>o</sup> | | | | X | X | X | X | X | $(X)^b$ | (X) | (X) <sup>b</sup> | |
| PROs <sup>p</sup> | (X) <sup>q</sup> | | (X) | (X) <sup>q</sup> | $(X)^q$ | (X) <sup>q</sup> | (X) <sup>q</sup> | X | $(X)^q$ | $(X)^q$ | $(X)^q$ | X |

Continued on Next Page

#### Continued

- \* The screening visit coincides with the end of study visit of the previous BAX855 study. The procedures/assessments marked with an asterisk (\*) will be transcribed from the end of study visit of the previous BAX855 study.
- Subjects transitioning from another BAX 855 study may have to repeat the PK assessment if evaluated to be necessary by the sponsor. The washout period prior to the PK determination is 72 96 hours, depending on the FVIII concentrate. PK will also be assessed at the 9-month visit (steady state PK) with the same post-infusion sampling timepoints.
- If a subject has a bleeding episode, instead of a phone visit the subject must attend a site visit to assess FVIII trough levels and IR and re-evaluate the PK-guided regimen (see Figure 2). In these cases the subject will undergo all planned assessments for a study visit, including assessment of vital signs, physical examination, and all laboratory assessments excluding clinical chemistry and the lipid panel.
- <sup>c</sup> Including subjects who withdraw or discontinue.
- d Occurs at enrollment (prior to any study-specific procedure).
  - <sup>e</sup> Medical history to include hemophilia history (confirmation of diagnosis & severity; family history of hemophilia; documentation of a mutation, if known; presence of any target joints; and historical ABR, blood group if available). Medication history to include documentation of all FVIII replacement therapies used within the last year, any prior history of use of any pegylated medication (eg, PEG-interferon) at any time in the past, and other medications in the last 30 days.
- Indicates that adverse events, concomitant medications, non-drug therapies, bleeding episodes and their treatment as well as the physical activity levels 8 hours prior to the occurrence of bleeding will be continuously monitored but specifically discussed and reviewed at these time points.
- Includes height and weight at screening, weight at the pre-infusion assessments, and Karnofsky performance score at screening.
- Pulse, respiration, supine blood pressure, and temperature to be assessed within 15 minutes prior to start of infusion and 30±5 minutes following infusion.
- The physical activity level in the 8 hours before the start of the bleeding episode should also be recorded.
- A target joint is defined as one in which there have been  $\geq 4$  bleeds in any consecutive 6-month period.
- The subject diary will be handed out at screening and training will be provided at the subsequent visits and the entries are reviewed and discussed with subject. It will be used to document bleeds, physical activity in the 8 hours before the bleed, treatment administered and response to BAX 855, prophylactic infusions, untoward events, concomitant medications, PROs and health resource use data, if applicable.
- For laboratory assessments, See Section 21.4.
- BAX 855 is administered in the clinic at the visits shown. At the PK assessment and for IR determination a set dose of  $60 \pm 5$  IU/kg BAX 855 is used, in all other cases the dose is PK-guided according to the allocated regimen.
- Transitioning subjects will receive IP of study 261303 as of the screening visit. Newly recruited subjects will continue with their previous treatment regimen until the first prophylactic PK guided infusion at baseline and the infusion for PK determination.
- In the first 6-month period, adjustments can be made based on PK and FVIII trough levels from previous study visits. Dose adjustments in second 6-month period are only permitted when FVIII trough levels are outside of the target window. Adjustments should be based on PK, pre-dose FVIII trough level from previous visit, any change in body weight, and assessment of any spontaneous bleeds. Before any dose adjustments are performed an additional visit should be scheduled within 14 days after receipt of FVIII activity results. Details of dose adjustments will be provided in a separate document.
- PROs include: Haemo-SYM Questionnaire, EQ-5D questionnaire, Short-Form 36 (SF-36), Physical Activity, and Health Resource Use; PROs can be done either at screening visit or baseline visit. Should always be completed before any study visit specific procedure.
- <sup>q</sup> EQ-5D, Patient Activity Level and Health Resource Use will be determined at each study visit.

# **21.4 Clinical Laboratory Assessments**

| | it | PK<br>Assessment <sup>b</sup> | Study Visits <sup>c</sup> | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures/<br>Assessments <sup>a</sup> | Screening Visit | Pre Infusion,<br>1530 Min,<br>3±0.5 h, 9±0.5 h,<br>32±2 h, 56±4 h<br>& 96±4 h<br>Post-Infusion | Baseline Visit | Visit<br>4Wk<br>±5d | Visit<br>8Wk<br>±1Wk | Visit<br>3 Mo<br>± 2Wk | Visit<br>4.5 Mo<br>±2Wk | Visit<br>6 Mo<br>±2Wk | Visit<br>7.5 Mo<br>±2Wk <sup>q</sup> | Visit<br>9 Mo<br>±2Wk<br>+PK | Visit<br>10.5 Mo<br>±2Wk <sup>q</sup> | Completion/<br>Termination<br>Visit <sup>d</sup> 12 Mo<br>±2Wk |
| Washout for FVIII and immunogenicity testing | None | 72-96 h | | | | days) or 8 | 84 hours ( | 3.5 day ii | itervals); | | gh arm: at | ter the short<br>least 48 h, or |
| CD4 count <sup>e</sup> | X | | | | | | | | | | | |
| Genetics and HLA-genotype <sup>f</sup> | X | | | | | | | | | | | |
| Viral serology <sup>g</sup> | X | | | | | | | | | | | |
| Blood type <sup>h</sup> | X | | | | | | | | | | | |
| Pregnancy Test (if applicable) <sup>i</sup> | X | | | | | | | | | | | |
| FVIII and<br>VWF:Ag assays <sup>j</sup> | X | X | $X^k$ | X | X | $X^k$ | X | $X^k$ | (X <sup>k</sup> ) | $X^k$ | (X <sup>k</sup> ) | $X^k$ |
| Immunogenicity <sup>l</sup> | X | | X | X | X | X | X | X | (X) | X | (X) | X |
| Hematology <sup>m</sup> | X | | X | | | X | | X | (X) | X | (X) | X |
| Clinical chemistry and lipid panel <sup>n</sup> | X | | X | | | X | | X | | X | | X |
| TGA° | X | X | X | X | X | X | X | X | (X) | X | (X) | X |
| Additional blood draw for further exploratory testing <sup>p</sup> | | | X | | | X | | | | X | | X |

Continued on Next Page

#### Continued

- At all assessments subjects must not be actively bleeding. In addition to the assessments shown, clinical laboratory tests should be performed whenever clinically indicated.
- Subjects transitioning from another BAX 855 study may have to repeat the initial PK assessment if evaluated to be necessary by the sponsor. The wash-out period prior to the PK determination is 72 96 hours, depending on the FVIII concentrate. PK will also be assessed at the 9-month visit (steady state PK) with the same post-infusion sampling timepoints.
- If a subject has a bleeding episode since the last visit before the 7.5 month ± 2 week or 10.5 month ± 2 week visits, instead of a phone visit the subject must attend a site visit to assess FVIII trough levels and IR and re-evaluate the PK-guided regimen. In these cases, the subject will undergo all assessments as listed for the 3 and 6 month ± 2 week visits.
- Including subjects who withdraw or discontinue.
- <sup>e</sup> CD4 count is analyzed in HIV positive subjects only to determine eligibility.
- If results of FVIII gene mutation analysis and HLA genotype are already available at the study site, they will be provided to the sponsor and an additional analysis will not be required.
- <sup>g</sup> Viral serology includes: HIV-1, HIV-2, HBcAb, HBsAb, HBsAg, HCVAb. Any HCV positive sample will be tested by PCR for viral titer.
- h If historical data on blood group type is available, this may be recorded in the CRF and blood type does not need to be determined.
- Pregnancy test as appropriate (serum pregnancy test in females of child-bearing potential if no urine sample is available). The pregnancy test might be repeated during the study in countries where mandated by national law.
- Factor VIII assays include: 1-stage clotting FVIII activity, FVIII chromogenic activity, and FVIII antigen. For assessment of trough levels, a blood sample will be taken within 30 minutes before the IP infusion. VWF antigen level will only be determined pre-infusion at each study visit.
- For assessment of FVIII IR, in addition to the pre-infusion sample a second sample will be taken 15-30 minutes after IP infusion.
- Immunogenicity assessments include: inhibitory antibodies to FVIII, binding antibodies to FVIII, BAX 855 and PEG, and anti-CHO antibodies. Both IgG and IgM binding antibodies will be measured. Blood draws have to be performed within 30 min before the IP infusion.
- <sup>m</sup> Hematology assessments include: hemoglobin, hematocrit, red blood cell count, and white blood cell count with differential (ie, basophils, eosinophils, lymphocytes, monocytes, and neutrophils), mean corpuscular volume (MCV), mean corpuscular hemoglobin concentration (MCHC), and platelet count. Samples should be taken within 30 minutes before the start of IP infusion.
- <sup>n</sup> Clinical chemistry assessments include: sodium, potassium, chloride, bicarbonate, total protein, albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, blood urea nitrogen (BUN), creatinine, and glucose. Lipid panel includes cholesterol, very low density lipoprotein (VLDL), low density lipoprotein (LDL), high density lipoprotein (HDL), and triglycerides. Samples should be taken within 30 minutes before the start of IP infusion.
- TGA parameters are lag time, time to peak thrombin generation, peak thrombin generation, and endogenous thrombin potential [ETP] Samples will be taken together with blood samples for FVIII activity and antigen determination.
- Blood draws for additional exploratory testing will be drawn pre-infusion and early in the morning if feasible, otherwise at the same time point at each study visit.
- <sup>q</sup> Only applicable for subjects who experience bleeding episodes since the previous study visit have to perform a study site visit.

#### 22. PERIOPERATIVE MANAGEMENT

# 22.1 Dosing Schedule and requirements for major surgery

#### **22.1.1** General

The dose and frequency of BAX 855 administered will be individualized based on the subject's IR and half-life, if available, and the required FVIII target levels.

The required units will be calculated according to the following formula:

Required units (IU) =

body weight (kg) x desired FVIII rise (IU/dL) x {reciprocal of IR} (IU/kg)/(IU/dL)

Example: In case of an IR of 2.0 [IU/dL]/[IU/kg], the required units would be calculated using the following formula:

body weight (kg) x desired FVIII rise (IU/dL) x 0.5 (IU/kg)/(IU/dL)

If at any time during the study, a subject does not respond to BAX 855 therapy as anticipated either by the operating surgeon or hemophilia physician providing postoperative care, blood samples will be drawn for the determination of FVIII activity levels and inhibitory antibodies to FVIII. In the event of unexplained, excessive bleeding, the subject will be treated by whatever means necessary until adequate hemostasis is achieved. The use of adjunct antifibrinolytic therapy such as e.g. tranexamic acid is allowed if clinically indicated by the investigator and/or according to the standard of care of the subject's institution.

# 22.1.2 Preoperative and Loading Dose

The subject will receive a loading dose calculated according to the formula described above in order to maintain a minimum target FVIII level as required by the category and type of surgery. The recommended loading dose will be calculated by the investigator.

The initial loading dose will be administered within 60 minutes prior to surgery (prior to incision/intubation). Vials of varying potencies may be used to ensure adequate dosing. A blood sample for post infusion FVIII at  $15 \pm 5$  minutes after completion of the initial loading dose will be drawn to ensure that the required FVIII levels have been obtained. Also, pre-infusion blood sample may be drawn within 30 minutes prior to the loading dose. Activated partial thromboplastin time (aPTT) will also be determined from the post infusion blood sample.

In case of major surgery, FVIII target levels should be 80-100% of normal, in case of minor surgery FVIII levels should be at 30 - 60%.

If the FVIII activity results are not available within a reasonable time period prior to the start of surgery, at least the post-infusion value of the aPTT must be obtained. The FVIII activity level following the loading dose must be obtained within 4 hours of infusion of BAX 855 and dose adjustments must be performed as needed.

# The surgery may only start after normalization of the aPTT.

If the aPTT is not normalized or the desired FVIII activity is not attained, a supplemental loading dose(s) of BAX 855 can be given at the discretion of the investigator.

Subsequent infusions of BAX 855 should be preceded by measurement of residual FVIII levels and dose adjustments must be based on the most recent residual FVIII activity levels.

# 22.1.3 Postoperative Dosing

After the initial loading dose, an optional re-bolus sufficient to raise FVIII levels to the appropriate level as defined for the type of surgery may be administered after a blood sample for FVIII determination has been drawn and the required FVIII levels by the local laboratory have been determined.

#### Note:

A second FVIII activity level should be determined within preferably 6-8 h following major surgery and within 12 h at the latest, with dose adjustments as necessary on the day of surgery.

ALL subsequent infusions of BAX 855 should be preceded by measurement of residual FVIII levels and the dose adjusted as needed. Dosing adjustments based on aPTT values are not allowed. Based on each individual PK parameters, ie, IR and half-life, if available, it is recommended that the following FVIII trough levels should be targeted for major surgery:

- The first postoperative 72 hours (Day 1- Day 3):  $\geq 80\%$
- Postoperative Day  $4 \text{Day } 7: \ge 50\%$  (if not yet discharged)
- Postoperative Day 8 to discharge (if not yet discharged): it is recommended that the FVIII levels should not fall below 30% (left to the discretion of the investigator depending on the postoperative course)

General postoperative treatment recommendations:

- Treatment intervals should be tailored in order not to exceed supraphysiological peak FVIII levels of 180%. Therefore, the dose should be administered in 1-3 infusions over 24 hours, most commonly in 2 infusions.
- The dose may be increased to a maximum of 100 IU/kg, however, the peak level should not exceed 180%.

Beginning postoperative Day 1 (ie, the day following the day of surgery) through discharge, subjects will have a BAX 855 pre-infusion (within 30 minutes) and after  $15\pm 5$  minutes a post-infusion FVIII level measurement at least once per day in order to assess the adequacy of factor replacement therapy during the postoperative period. For consistency, it is recommended that the daily blood draws are performed at the same time of the day, eg, morning blood draws. At a minimum, a blood sample for FVIII determination must be drawn prior to any supplemental unscheduled FVIII infusion.

Figure 3 is a visualization of timing and target FVIII levels for major surgery.



Figure 3
Dosing Recommendations for Major Surgeries

# 22.2 Efficacy assessment

# 22.2.1 Intra-, Post-, and Perioperative Hemostatic Efficacy

The hemostatic efficacy will be assessed during (Table 5) and after (Table 6) any surgical or invasive procedures, and overall as a perioperative assessment (Table 7).

| | Table 5 Intraoperative Efficacy Assessment Scale | |
|---|---|---|
| | Prior to the discharge from the recovery room, the operating surgeon will assess the intraoperative hemostatic efficacy compared to that expected for the type of procedure performed in a non-hemophilic population | |
| Rating | Criteria | Score |
| Excellent | Intraoperative blood loss was less than or equal to that expected (≤100%) | 3 |
| Good | Intraoperative blood loss was up to 50% more than expected (101-150%) | 2 |
| Fair | Intraoperative blood loss was more than 50% of that expected (>150%) | 1 |
| None | Uncontrolled hemorrhage that was the result of inadequate therapeutic response despite proper dosing, necessitating rescue therapy | 0 |

| | Table 6 Postoperative Efficacy Assessment Scale (Postoperative Day 1) | |
|---|---|---|
| | On postoperative Day 1, the operating surgeon will assess the postoperative hemostatic efficacy compared to that expected for the type of procedure performed in a non-hemopopulation | |
| Rating | Criteria | Score |
| Excellent | Postoperative blood loss was less than or equal to (≤100%) that expected | 3 |
| Good | Postoperative blood loss was up to 50% more (101-150%) than expected | 2 |
| Fair | Postoperative blood loss was more than 50% (>150%) of that expected | 1 |
| None | Significant postoperative bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating rescue therapy | 0 |

| Perio | Table 7<br>perative Efficacy Assessment Scale (at discharge or 14 days post-surgo<br>whichever is first) | ery, |
|---|---|---|
| | At discharge or 14 days post-surgery, whichever is first, a hematologist will assess the perioperative efficacy compared to that expected for the type of procedure performed in hemophilic population | n a non- |
| Rating | Criteria | Score |
| Excellent | Perioperative blood loss was less than or equal to (≤100%) that expected Required blood components for transfusions were less than or similar to that expected | 3 |
| Good | Perioperative blood loss was up to 50% more (101-150%) than expected Required blood components for transfusions were less than or similar to that expected | 2 |
| Fair | Perioperative blood loss was more than 50% of that expected (>150%) Required blood components transfusions were greater than that expected | 1 |
| None | Significant perioperative bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating rescue therapy Required blood components for transfusions were substantially greater than expected | 0 |

# 22.2.2 Intra- and Postoperative Blood Loss

The observed versus predicted operative blood loss will be described for the period from initiation of the intervention to discharge or 14 days after the intervention, whichever is first.

Prior to the surgery, the surgeon/investigator will predict the estimated volume (mL) of the expected average and maximum blood loss for the planned surgical intervention in a hemostatically normal individual of the same sex, age, and stature as the study subject, for intraoperative, postoperative and overall perioperative time periods. Every effort should be made to predict the volume as precisely as possible, also taking into account, for example, the use of a tourniquet or placement of a postoperative drain and whether or not suction is used. The estimate will be for the intraoperative time period from completion of the procedure until approximately 24 hours post-surgery and for the overall perioperative time period (assessed at discharge or 14 days after the intervention, whichever is first).

The intraoperative blood loss will be measured by determining the volume of blood and fluid removal through suction into the collection container (waste box and/or cell saver) and the estimated blood loss into swabs and towels during the procedure, per the anesthesiologist's record. Post-operatively, blood loss will be determined by the drainage volume collected, which will mainly consist of drainage fluid via vacuum or gravity drain, as applicable. In cases where no drain is present, blood loss will be determined by the surgeon's clinical judgment, as applicable or entered as "not available".

#### 23. DEFINITIONS

#### 23.1 Joint Bleeds

Features of an acute joint bleed include some or all of the following: 'aura', pain, swelling, warmth of the skin over the joint, decreased range of motion and difficulty in using the limb compared with baseline or loss of function.

The earliest clinical signs of a joint bleed are increased warmth over the area and discomfort with movement, particularly at the ends of range.

Later symptoms and signs include pain at rest, swelling, tenderness, and extreme loss of motion.

In patients with advanced arthropathy it may be difficult to distinguish pain-related arthritis from that associated with an acute bleed. Rapid resolution of pain following infusion of factor concentrates (typical of an acute hemarthrosis) or improvement of pain associated with activity soon after a period of rest (typical of chronic arthritis) can help distinguish between the two.

In infants and young children, reluctance to use the limb alone may be indicative of a joint/muscle bleed.

#### 23.2 Muscle Bleeds

Muscle bleeds can occur in any muscle of the body, usually from a direct blow or a sudden stretch. A muscle bleed is defined as an episode of bleeding into a muscle, determined clinically and/or by imaging studies, generally associated with pain and/or swelling and functional impairment over baseline.

For further definitions of CNS, GI and abdominal hemorrhages see the Guidelines for the management of hemophilia from the world federation of hemophilia. 31;32

#### 24. REFERENCES

- 1. Björkman S, Berntorp E. Pharmacokinetics of coagulation factors: clinical relevance for patients with haemophilia. Clin.Pharmacokinet. 2001;40:815-832.
- 2. Björkman S, Folkesson A, Jönsson S. Pharmacokinetics and dose requirements of factor VIII over the age range 3-74 years: A population analysis based on 50 patients with long-term prophylactic treatment for haemophilia A. Eur.J.Clin.Pharmacol. 2009;65:989-998.
- 3. Valentino, L. A., Mamonov, V., Hellmann, A., Quon, D., Desmond, J. C., Schroth, P., and Wong, W. Y. Prophylaxis in haemophilia A: A multicenter, open-label, randomized, phase 4 clinical study of ADVATE. 2011.
- 4. White GC, II, Rosendaal F, Aledort LM et al. Definitions in hemophilia. Recommendation of the scientific subcommittee on factor VIII and factor IX of the scientific and standardization committee of the International Society on Thrombosis and Haemostasis. Thromb.Haemost. 2001;85:560-575.
- 5. Boggio LN, Kessler CM. Hemophilia A and B. In: Kitchens C, Alving B, Kessler C, eds. Consultative Hemostasis and Thrombosis. Philadelphia: Saunders Elsevier; 2007:43, 45-59.
- Committee for Medicinal Products for Human Use. Guideline on the clinical investigation of recombinant and human plasma-derived factor VIII products. EMA/CHMP/BPWP/144533/2009. 7-21-2011. European Medicines Agency (EMA).

Link to Publisher's Site:

http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/201 1/08/WC500109692.pdf

- 7. Acharya SS: Exploration of the pathogenesis of haemophilic joint arthropathy: understanding implications for optimal clinical management. Br.J.Haematol. In press.
- 8. Valentino LA. Blood-induced joint disease: the pathophysiology of hemophilic arthropathy. J.Thromb.Haemost. 2010;8:1895-1902.
- 9. Blanchette VS, Manco-Johnson M, Santagostino E, Ljungs R. Optimizing factor prophylaxis for the haemophilia population: where do we stand? Haemophilia. 2004;10 Suppl 4:97-104.
- Manco-Johnson M. Comparing prophylaxis with episodic treatment in haemophilia
   A: implications for clinical practice. Haemophilia. 2007;13 Suppl 2:4-9.
- 11. Gringeri A, Bianchi B. Evaluation study on prophylaxis: A randomised italian trial (ESPRIT). One-Year Report [abstract]. Haemophilia. 1998;4:171.
- 12. Gringeri A. Evaluation study on prophylaxis: a randomised Italian trial (Esprit). two-years report [abstract]. 1999;
- 13. Fischer K. Can we consider discontinuing primary prophylaxis in adults with severe haemophilia? Haemophilia. 2008;14 Suppl 4:10.
- 14. Fischer K, van der Bom JG, Mauser-Bunschoten EP et al. Changes in treatment strategies for severe haemophilia over the last 3 decades: effects on clotting factor consumption and arthropathy. Haemophilia. 2001;7:446-452.
- 15. Fischer K, van der Bom JG, Negrier C, Grobbee DE, van den Berg M. Comparing Prophylaxis to on Demand Treatment for Severe Hemophilia: Better Outcome at Equal Costs [abstract]. Blood. 2001;98 Suppl 1:533a.
- 16. Fischer K, Astermark J, van der Bom JG et al. Comparison of the two prophylactic regimens for severe hemophilia: Intermediate dose versus high dose [abstract]. Blood. 2001;98 Suppl 1:532a.

- 17. Manco-Johnson M, Abshire T, Brown D et al. Initial results of a randomized, prospective trial of prophylaxis to prevent joint disease in young children with factor VIII (FVIII) deficiency [abstract]. Blood. 2005;106:6a.
- Gringeri A, Lundin B, von Mackensen S et al. A randomized clinical trial of prophylaxis in children with hemophilia A (the ESPRIT Study).
   J.Thromb.Haemost. 2011;9:700-710.
- National Hemophilia Foundation. Recommendation concerning prophylaxis (Prophylactic administration of clotting factor concentrate to prevent bleeding).
   MASAC 117. 5-19-2001. National Hemophilia Foundation (NSF).
- National Hemophilia Foundation. Recommendation Concerning Prophylaxis (Regular Administration of Clotting Factor Concentrate to Prevent Bleeding).
   MASAC 170. 4-22-2006. National Hemophilia Foundation (NHF).
- 21. National Hemophilia Foundation. Recommendation concerning prophylaxis (Regular administration of clotting factor concentrate to prevent bleeding). MASAC 179. 4-11-2007. National Hemophilia Foundation (NHF). Link to Publisher's Site: https://www.hemophilia.org/sites/default/files/document/files/masac179.pdf
- 22. Ahnström J, Berntorp E, Lindvall K, Björkman S. A 6-year follow-up of dosing, coagulation factor levels and bleedings in relation to joint status in the prophylactic treatment of haemophilia. Haemophilia. 2004;10:689-697.
- 23. den Uijl IEM, Mauser Bunchoten EP, Roosendaal G et al. Clinical severity of haemophilia A: does the classification of the 1950s still stand? Haemophilia. 2011;17:849-853.
- 24. Funk M, Schmidt H, Escuriola-Ettingshausen C et al. Radiological and orthopedic score in pediatric hemophilic patients with early and late prophylaxis.

  Ann.Hematol. 1998;77:171-174.

25. Funk MB, Schmidt H, Becker S et al. Modified magnetic resonance imaging score compared with orthopaedic and radiological scores for the evaluation of haemophilic arthropathy. Haemophilia. 2002;8:98-103.

Page 106 of 110

2015 MAY 12

- 26. Lundin B, Ljung R, Pettersson H, The European Paediatric Network for Haemophilia Management (PEDNET). MRI scores of ankle joints in children with haemophilia comparison with clinical data. Haemophilia. 2005;11:116-122.
- Aledort LM, Haschmeyer RH, Pettersson H. A longitudinal study of orthopaedic outcomes for severe factor-VIII-deficient haemophiliacs. The Orthopaedic Outcome Study Group. J.Intern.Med. 1994;236:391-399.
- 28. Nilsson IM, Berntorp E, Lofqvist T, Pettersson H. Twenty-five years' experience of prophylactic treatment in severe haemophilia A and B. J.Intern.Med. 1992;232:25-32.
- 29. van Dijk K, Fischer K, van der Bom JG, Grobbee DE, van den Berg HM. Variability in clinical phenotype of severe haemophilia: the role of the first joint bleed. Haemophilia. 2005;11:438-443.
- 30. Feldman BM, Funk SM, Bergstrom BM et al. Validation of a new pediatric joint scoring system from the international hemophilia prophylaxis study group: Validity of the hemophilia joint health score (HJHS). Arthritis Care Res. 2011;63:223-230.
- 31. Blanchette VS, Key NS, Ljung LR et al. Definitions in hemophilia: Communication from the SSC of the ISTH. J.Thromb.Haemost. 2014;12:1935-1939.
- 32. World Federation of Hemophilia Treatment Guidelines Working Group and Srivastava, A. Guidelines for the management of hemophilia 2nd Edtion. 2005. World Federation of Hemophilia (WFH).

  Link to Publisher's Site: http://www1.wfh.org/publication/files/pdf-1472.pdf

#### 25. SUMMARY OF CHANGES

Protocol 261303: Amendment 2 2015 MAY 12 Replaces: Amendment 1 2015 MAR 20

In this section, changes from the previous version of **Amendment 1**, dated **2015 MAR 20**, are described and their rationale is given.

# 1. Throughout the document.

<u>Description of Change</u>: The term PEG written in capital letters for example "PEGylation" and "PEGylated" was changed to lower case letters "pegylation" and "pegylated". Minor grammatical and/or administrative changes have been made.

<u>Purpose for Change</u>: To be consistent with internal guidelines and to improve the readability and/or clarity of the protocol.

2. Sections: Synopsis, 6.4.2 Finding from Clinical Studies, 7.3.4 Patient Reported Outcomes, 7.4 Exploratory Objectives, 8.4.2.3 Patient Reported Outcomes, 8.4.3 Exploratory Outcome Measures, 14.4.2 Secondary Outcome Measures, 14.4.3 Exploratory Outcome Measures

<u>Description of Change</u>: Details on Patient Reported Outcomes and their use for assessment of secondary outcome measures were added

<u>Purpose for Change</u>: To provide additional information

3. Sections: Synopsis, 7.3.1 Objectives - Efficacy, 8.4.2.1 Outcome Measures - Efficacy, 8.7.3.5 Treatment for Surgery or Dental procedures, 9.2 Exclusion Criteria 9.3 Withdrawal and Discontinuation 10.4 Medications and Non-Drug Therapies 11.1.5 Perioperative Efficacy Assessments 14.4.1 Primary Outcome Measure 14.4.2 Secondary Outcome Measures 22 Supplement: Perioperative Management

# Description of Change:

A surgery arm was included in the study protocol. Details for perioperative management are provided in the supplement. The necessary revisions are made throughout the protocol.

<u>Purpose for Change</u>: Surgeries are now in the scope of this study to avoid potential drop-outs in case major surgeries are required and the surgery protocol (study protocol 261204) is not in place.

4. Sections: Synopsis, 14.1.1 Sample Size Calculation, 14.3 Handling of Missing, Unused and Spurious Data, 14.3.2 Handling of other variables, 14.4.1 Primary Outcome Measure, 14.4.2 Secondary Outcome Measures, 14.5 Planned Interim Analysis of the Study.

# Description of Change:

Details in statistical analysis were added:

- a) Specifications for the handling of missing data, including assumptions how missing data will be used for the analysis methods and a plan for sensitivity analyses to assess the impact of assumptions regarding the missing data mechanism of the analysis results.
- b) Subgroup analyses with respect to age and race will be included
- c) The Chi-squared test with continuity correction is used which results in a lower but acceptable power of 80%.
- d) The section for the planned interim analysis was deleted
- e) Definition of the interruption period in case of surgery. Description how the secondary outcome measures related to surgical procedures will be analyzed.

# <u>Purpose for Change</u>:

- a) and b) Upon regulatory request
- c) To account for a more conservative approach considering continuity correction.
- d) A planned interim analysis will not be performed.
- e) To account for the surgical procedures.

# 5. Section 8.5 Randomization and blinding

<u>Description of change</u>: The following sentence was added: Randomization occurs after the PK assessment and will be stratified according to subjects' pre-study treatment regimen (prophylaxis vs. on-demand).

<u>Purpose for change</u>: To account for pretreatment regimen.

# 6. Sections: 12.1 Pharmacokinetics, 21.2 Detailed Flow Diagram of Study Procedures, 21.3 Schedule of Study Procedure and Assessments, 21.4 Clinical Laboratory Assessments

# <u>Description of Change</u>:

The blood sampling time points for PK study were modified as follows: Post-infusion at 15-30 minutes and at 3, 8, 24, 48, 72 and 96 hours.

Purpose for Change: Upon regulatory request.

# 7. Sections: 8.7.3.3 BAX 855 Dose and/or Frequency Adjustments 12.3 Trough Levels, 21.3 Schedule of Study Procedures and Assessments

# Description of Change:

A repeat FVIII trough level measurement will be performed approximately 2 weeks after dose adjustment.

# Purpose for Change:

Upon regulatory request: to ensure that the adjusted dose is adequate. After approximately 2 weeks the subject will have reached steady state.

# 8. Section 8.7.3.4 Treatment of bleeding episodes

<u>Description of change</u>: The dose calculation for treatment of bleeding episodes was revised.

Purpose for change: Inadvertently, FIX was written instead of FVIII.

#### INVESTIGATOR ACKNOWLEDGEMENT

# BAX 855 - Pegylated Full-Length Recombinant Factor VIII

Phase 3, prospective, randomized, multi-center clinical study comparing the safety and efficacy of BAX 855 following PK-guided prophylaxis targeting two different FVIII trough levels in subjects with severe Hemophilia A

**PROTOCOL IDENTIFIER: 261303** 

**CLINICAL TRIAL PHASE 3** 

AMENDMENT 2: 2015 MAY 12 Replaces: AMENDMENT 1: 2015 MAR 20

ALL VERSIONS:

AMENDMENT 2: 2015 MAY 12 AMENDMENT 1: 2015 MAR 20 ORIGINAL: 2015 JAN 13

# OTHER ID(s)

NCT Number: To be Determined

EudraCT Number: To be Determined

IND NUMBER: To be Determined

By signing below, the investigator acknowledges that he/she has read and understands this protocol, and provides assurance that this study will be conducted according to all requirements as defined in this protocol, clinical study agreement, ICH GCP guidelines, and all applicable regulatory requirements.

| Signature of Coordinating Investigator | | Date | |
|----------------------------------------|----------------------|------|----|
| Print Name and Title of Coord | inating Investigator | | - |
| ia. | | | |
| Signature of Sponsor Represen | ıtative | Date | 93 |